

# **Non-interventional Study Protocol**

| Document Number: | 1.0 |
|---|---|
| BI Study Number: | 1160.253 |
| BI Investigational Product(s): | Dabigatran etexilate (Pradaxa®) |
| Title: | Non-interventional study describing treatment convenience in patients treated with Dabigatran for Stroke Prophylaxis in Atrial Fibrillation (SPAF) |
| Protocol version identifier: | Final 1.0 |
| Date of last version of protocol: | 30 Nov 2015 |
| PASS: | No |
| EU PAS register<br>number: | N.A. |
| Active substance: | Anatomical main group: B - Blood and blood forming organs Therapeutic subgroup: B01 - Antithrombotic agents Pharmacological subgroup: B01A - Antithrombotic agents Chemical subgroup: B01AE - Direct thrombin inhibitors Chemical substance: B01AE07 - Dabigatran etexilate. |
| Medicinal product: | Dabigatran etexilate |
| Product reference: | EU/1/08/442. |
| Procedure number: | EMEA/H/C/829 |
| Marketing authorisation holder(s): | Boehringer Ingelheim International GmbH<br>Binger Str. 173<br>D-55216 Ingelheim am Rhein<br>Germany |
| Joint PASS: | No |

| Research question and objectives: | Primary objective: Describe the atrial fibrillation patient's treatment perception by using the PACTQ-2 at three time-points at baseline, during initiation period and during the continuation period. |
|---|---|
|---|---|

| Secondary objective: | |
|---|---|
| | Characterization of patient population (including dosing) in Spain. |
| Country(-ies) of study: | Spain |
| Author: | |
| | Tel:<br>Fax:<br>Mobile: |
| Marketing authorisation holder(s): | Boehringer Ingelheim International GmbH<br>Binger Str. 173<br>D-55216 Ingelheim am Rhein<br>Germany |
| MAH contact person: | Not applicable |
| EU-QPPV: | Not applicable |
| Signature of EU-QPPV: | Not applicable |
| Date: | 30 Nov 2015 |

**Proprietary confidential information** 

© 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

# 1. TABLE OF CONTENTS

| 1. | TABL | E OF CONTENTS | 3 |
|---|---|---|---|
| 2. | LIST C | OF ABBREVIATIONS | 5 |
| 3. | RESPO | ONSIBLE PARTIES | 6 |
| 4. | ABSTI | RACT | 7 |
| 5. | AMEN | IDMENTS AND UPDATES | 11 |
| 6. | MILES | STONES | 12 |
| 7. | RATIO | NALE AND BACKGROUND | 13 |
| 8. | RESEA | ARCH QUESTION AND OBJECTIVES | 14 |
| 8.1 | RES | SEARCH QUESTIONS | 14 |
| 8.2 | OB. | JECTIVES: | 14 |
| 9. | RESEA | ARCH METHODS | 15 |
| 9.1 | STU | JDY DESIGN | 15 |
| 9.2 | SET | TING | 15 |
| 9 | .2.1 | Selection of sites: | 15 |
| 9 | .2.2 | Inclusion criteria: | 16 |
| 9 | .2.3 | Exclusion criteria: | 16 |
| 9 | .2.4 | Removal of patients from the study | 16 |
| 9 | .2.5 | Visit schedule | |
| 9 | .2.6 | Treatments | |
| 9 | .2.7 | Concomitant medications and restrictions | |
| 9 | .2.8 | Representativeness of the study population: | |
| 9.4 | | RIABLES | |
| | .4.1 | Primary objective: | |
| | | For Secondary objectives | |
| 9.5 | | ΓA SOURCES | |
| 9.6 | | JDY SIZE | |
| 9.7 | | ΓΑ MANAGEMENT | |
| 9.8 | | FA ANALYSIS | |
| _ | .8.1 | STUDY DESIGNPLANNED ANALYSES | |
| 9 | .8.2<br>9.8.2.1 | | |
| | 9.8.2.1 | • | |
| | | Safety Analyses Safety Analyses | |
| | 1.0.4 | / Duicty / High voca | <i></i> / |

| 9.8.2.4 Schedule of Planned Analyses | 27 |
|--------------------------------------------------------------------|------|
| 9.8.3 HANDLING OF MISSING DATA | 28 |
| 9.9 QUALITY CONTROL | 28 |
| 9.10 LIMITATIONS OF THE RESEARCH METHODS | 28 |
| 9.11 OTHER ASPECTS | 30 |
| 9.11.1 INFORMED CONSENT, DATA PROTECTION, STUDY RECORD | )S30 |
| 9.11.1.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT | 30 |
| 9.11.1.2 DATA QUALITY ASSURANCE | 30 |
| 9.11.1.3 RECORDS | |
| 9.11.1.3.1 Source documents | 31 |
| 9.11.1.3.2 Direct access to source data and documents | 31 |
| 9.11.1.4 STATEMENT OF CONFIDENTIALITY | 31 |
| 9.11.1.5 COMPLETION OF STUDY | 32 |
| 10. PROTECTION OF HUMAN SUBJECTS | 33 |
| 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | |
| 11.1 Definitions of adverse events | 34 |
| 11.2 Adverse event and serious adverse event reporting | 35 |
| 11.3 Time windows | 36 |
| 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY | |
| RESULTS | 37 |
| 13. REFERENCES | 38 |
| 13.1 PUBLISHED REFERENCES | 38 |
| 13.2 UNPUBLISHED REFERENCES | 39 |
| ANNEX 1. LIST OF STAND-ALONE DOCUMENTS | 40 |
| ANNEX 2. ENCEPP CECKLIST FOR STUDY PROTOCOLS | 48 |
| ANNEX 3 ADDITIONAL INFORMATION | 40 |

# 2. LIST OF ABBREVIATIONS

| AE | Adverse Event |
|---|---|
| AF | Atrial Fibrillation |
| ADR | Adverse Drug Reaction |
| BI | Boehringer Ingelheim |
| CA | Competent Authority |
| CHA <sub>2</sub> DS <sub>2</sub> - | Congestive heart failure, Hypertension, Age (> 75), |
| VASc score | Diabetes mellitus, Stroke/TIA, Vascular disease, Age 65-74, Sex |
| | Category |
| CI | Confidence Interval |
| CML | Local Clinical Monitor |
| CRA | Clinical Research Associate |
| CRF | Case Report Form |
| DMP | Data Management Plan |
| eCRF | Electronic Case Report Form |
| DEDP | Drug Exposure During Pregnancy |
| EC | Ethics Committee |
| ECG | Electrocardiogram |
| EDC | Electronic Data Capture |
| EMA | European Medicine Agency |
| EudraCT | European Clinical Trials Database |
| FDA | Food and Drug Administration |
| GPV CTC | Global Pharmacovigilance Clinical Trial Coordinator |
| HAS-BLED | Hypertension, Abnormal renal and liver function, Stroke (1 point), Bleeding history or predisposition, Labile INR, Elderly (>65 years), Drugs and Alcohol. |
| HRQoL | Health related Quality of Life |
| ICSR | Individual Case Safety Report |
| IEC | Independent Ethics Committee |
| INR | International Normalized Ratio |
| IRB | Institutional Review Board |
| ISF | Investigator Site File |
| OPU | Operative Unit |
| OAC | Oral anticoagulation |
| PACTQ | Perception of Anticoagulation Treatment Questionnaire |
| SAE | Serious Adverse Event |
| SDV | Source Data Verification |
| SEAP | Statistical and Epidemiological Analysis Plan |
| SmPC | Summary of Product Characteristics |
| SOP | Standard Operating Procedure |
| SPAF | Stroke Prophylaxis in Atrial Fibrillation |
| VKA | Vitamin K Antagonist |

# 3. RESPONSIBLE PARTIES

| Therapeutic Area Cardiovascular Medicine |
|------------------------------------------|
| Team Member Medical Affairs |
| Team Member Epidemiology |
| Trial Clinical Monitor |
| Trial Statistician |
| GPV CTC |
| LPVM |
| Coordinator Investigator |

# 4. ABSTRACT

| Name of company: Pradaxa® | | | |
|---|---|---|---|
| Name of company: Boehringer Ingelheim | | Dabigatran | |
| <u> </u> | | etexilate, | |
| Name of finished medicinal product: Dabigatran etexilate | | ctexitate, | |
| | Name of active ingredient: | | |
| Anatomical main group | | | |
| forming organs Therap | | | |
| Antithrombotic agents | | | |
| Pharmacological subgre | oup: B01A - Antithrombotic | | |
| agents | | | |
| Chemical subgroup: B( inhibitors | OTAE - Direct thrombin | | |
| Chemical substance: Bo | 01 A F 07 - Dahigatran | | |
| etexilate. | OTALO7 - Daoigatian | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision |
| 30 Nov 2015 | 1160.253 | Final 1.0 | date: n/a |
| Title of study: | Non-interventional study | , describing treatmen | t convenience in |
| Title of study. | patients treated with Dab | <u> </u> | |
| | Fibrillation (SPAF) | nganan ioi Shoke i i | opilylaxis ili Autai |
| B 4 1 1 | | | |
| Rationale and | | sm prevention in AF | patients requires |
| background: | anticoagulation | | |
| | • In EU many antico | agulation strategies | are used: mainly |
| | _ | | _ |
| | Vitamin K antagonists (VKA), antiplatelet treatment and new anticoagulation therapies such as Pradaxa® | | |
| | • Atrial Fibrillation (AF) treatment varies widely by | | |
| | objective information e.g. prescribing information and patient | | |
| | and physicians perception | | |
| | Decision for choice of anticoagulation therapy and dose<br>selection is based on physician factors and patient factors | | |
| | Study rationale: characterize non-valvular AF patients treated | | |
| | with any recent VKA therapy and now newly initiated on | | |
| | Pradaxa® (switch patien | 1.0 | |
| Dagaawah arrastiss | | | C 1: 11 |
| Research question and objectives: | Describe patient and phys | | |
| and objectives. | being when treated with I | | |
| | prevention in non-valvula | | ther compared to |
| | previous antithrombotic treatment (switcher) | | |
| | Primary research interest: | | |
| | Describe the non-valvular AF patient well-being by using the | | |
| | PACTQ-2 at three time-p | oints when (1) being | treated with any |
| | anticoagulation therapy to | prevent stroke/embo | olism and planned to |
| | be switched (baseline to c | 1 | |
| | (2) being initiated on Prac | - | <b>-</b> - / |
| | Pradaxa® (~180 days). | (2 2 2 4 4 4 4 5 ) 0 | (-) |
| | Secondary Research inter | est: | |
| | Secondary Research Inter | CSI. | |

| 1) Characterization of patient population (incl. dosing): |
|---|
| <ol> <li>Patient demographic (age, gender, comorbidities, comedication)</li> </ol> |
| 3) Physician rated items to calculate HAS-BLED risk assessment at baseline |
| 4) Physician rated items to calculate CHA2DS2-VASc score at baseline |
| 5) If available: laboratory assessment of kidney function and calculation of Creatinine Clearance using CG-Formula |
| 6) Initial Pradaxa® dosing |
| 7) Reasons for Pradaxa® dose change and Pradaxa®/VKA discontinuation |
| Prospective, non-interventional study of non-valvular AF patients in Spain with a current VKA therapy and subsequent initiation of Pradaxa®. The inclusion of the patient in the study is not related with the decision of dabigatran prescription. Dabigatran prescription is based in the Health authorities recommendations in the positiong report of NACOs |
| _ |

| Population: | Patients diagnosed with non-valvular atrial fibrillation and eligible for change from VKA to Pradaxa® treatment according to Pradaxa® Summary of Product Characteristics. The inclusion of the patient in the study is not related with the decision of dabigatran prescription. Dabigatran prescription is based in the Health authorities recommendations in the positiong report of NACOs |
|---|---|
| Variables: | For objective 1: |
| | Outcome 1: Mean PACT-Q2 scores at second and last assessment compared to baseline assessment. |
| | Outcome 2: Mean PACT-Q2 score at last assessment compared to second assessment. |
| | For objective 2: |
| | Outcome 1: Characterization of patients according to |
| | - Age |
| | - Gender |
| | - CHA <sub>2</sub> DS <sub>2</sub> -VASc score (R10-5332) |
| | - HAS-BLED score (R10-6394) |
| | - Kidney function (creatinine clearance) |
| | <ul> <li>Stroke and/or bleeding related risk factors in medical<br/>history and at baseline</li> </ul> |
| | - Concomitant diseases |
| | - Concomitant therapies |
| | - Dosing of Pradaxa® |
| | - Duration of previous VKA treatment |
| Data sources: | <ul> <li>Newly generated data from enrolled patients (electronic CRF):</li> <li>Patient characteristics completed by physician's judgement and records.</li> <li>Questionnaires completed by patients.</li> </ul> |
| | - Creatinine clearance for assessment of kidney function will be calculated within the eCRF, by entering Creatinine values (from existing lab reports, if available) |
| Study size: | Up to 1087 patients in Spain |
| Data analysis: | In this non-interventional study, cross-sectional data at study baseline and longitudinal follow-up data over 6 months will be collected for non-valvular AF patients with a current VKA therapy and subsequent initiation of Pradaxa®. Baseline data will be described using a cross-sectional approach. Data from the longitudinal follow-up will be summarized descriptively. |
| Milestones: | Start of data collection: Planned June 2016 |

## Boehringer Ingelheim Non-interventional Study Protocol BI Study Number 1160.253


| End of data collection: Planned June 2017 |
|-------------------------------------------------------|
| Final report of study results: Planned September 2017 |

# 5. AMENDMENTS AND UPDATES

None.

# 6. MILESTONES

| Milestone | Planned Date |
|-------------------------------------|----------------|
| Start of data collection | June 2016 |
| End of data collection | June 2017 |
| Registration in the EU PAS register | Not applicable |
| Final report of study results: | September 2017 |

## 7. RATIONALE AND BACKGROUND

Pradaxa® (Dabigatran etexilate) is a direct Thrombin inhibitor approved in Europe, USA and many other countries worldwide for the prevention of stroke and systemic embolism in adult patients with non-valvular atrial fibrillation with one or more risk factors.

Pradaxa® has been studied in the RE-LY study, one of the largest non-valvular atrial fibrillation outcome studies (<u>P13-05668</u>). Over the course of one year, all anticoagulated patients without outcome events (e.g. strokes or major bleedings) had stable HRQoL. Scores between dabigatran and warfarin were comparable, which was unexpected given the known complexities of warfarin treatment. Other data on how patients perceive Pradaxa® treatment in the context of non-valvular atrial fibrillation disease management only exist to a limited degree in Europe. (R15-1312)

It is the aim of this non-interventional study to describe the patient perception of anticoagulation with a current VKA therapy and subsequent initiation of treatment with Pradaxa® to prevent stroke and systemic embolism while suffering from non-valvular atrial fibrillation (according to its approved indication in the approved dosages of 110 mg or 150 mg twice daily). The inclusion of the patient in the study is not related with the decision of dabigatran prescription. Dabigatran prescription is based in the Health authorities recommendations in the positiong report of NACOs

To evaluate patient understanding of treatment and patient values it is important to assess patient's perception of the treatment in the context of overall disease management as close as possible to the clinical practice. Furthermore it is important to anchor these data either to perception about a previous anticoagulation therapy.

These real world data are needed to guide the scientific community in designing educational efforts for doctors and their patients and to assess the potential values of patient adherence programs when using Pradaxa® as the first novel anticoagulant. Also such data, describing patient's perception on Pradaxa® anticoagulation in the context of patient-physician interaction managing stroke prevention in non-valvular atrial fibrillation cannot be obtained by market research. Thus, this non-interventional study is the appropriate methodology to address this research question.

## 8. RESEARCH QUESTION AND OBJECTIVES

## 8.1 RESEARCH QUESTIONS

This non-interventional study will address the following questions:

- How do patients with non-valvular atrial fibrillation perceive anticoagulation treatment for stroke prevention (switched from previous treatment to Pradaxa®)?
- Is there any geographical variation (between autonomous communities) in treatment convenience?
- Is there a variation of treatment convenience and treatment satisfaction among different age groups?
- What are the characteristics of patients receiving anticoagulation treatment for stroke prevention regarding demographics, physician rated risk scores, kidney function, concomitant diseases and concomitant medications, treatment for SPAF (choice of treatment, dosing)?

#### **8.2 OBJECTIVES:**

## **Primary objective**

Describe the non-valvular atrial fibrillation patient's treatment perception by using the PACTQ at three time-points: at baseline, during initiation period and during the continuation period:

- At baseline: when being treated with any anticoagulation therapy to prevent stroke/embolism and switched (baseline to capture VKA treatment perception). The inclusion of the patient in the study is not related with the decision of dabigatran prescription. Dabigatran prescription is based in the Health authorities recommendations in the positiong report of NACOs
- Initiation period: when being initiated on Pradaxa® (30-45 days).
- Continuation period: when continued on Pradaxa® (~180 days).

## **Secondary objective**

Characterization of patient population (incl. dosing) in Spain:

- Patient demographic (age, gender, comorbidities, co-medication)
- Physician rated items to calculate HAS-BLED risk assessment at baseline
- Physician rated items to calculate CHA2DS2-VASc score at baseline
- If available: laboratory assessment of kidney function and calculation of Creatinine Clearance using CG-Formula
- Initial Pradaxa® dosing
- Reasons for Pradaxa® dose change and Pradaxa®/VKA discontinuation

## 9. RESEARCH METHODS

#### 9.1 STUDY DESIGN

This is a non-interventional national, multi-centre study based on newly collected data. The study will enrol consented patients with non-valvular atrial fibrillation in Spain with a VKA therapy and subsequent initiation of Pradaxa®

This is an observational study since Pradaxa is prescribed according to the usual clinical practice, based on the Health Authority's recommendations. The therapeutic strategy assigned to the patient will not be decided according to any clinical trial protocol, but it will be determined according to the usual clinical practice. The prescription of any drug will be completely dissociated from the decision to include the patient in the study. The patient should not receive any intervention, whether diagnostic or monitoring, other than the usual clinical practice.

Patients will be followed over an observation period of 6 months. Data will be collected at three time points:

- 1. At Baseline (initiation on Pradaxa®)
- 2. 30-45 days after initiation on Pradaxa® (initiation period)
- 3. 150-210 days after initiation on Pradaxa® (continuation period)

#### 9.2 SETTING

It is planned that data of approximately 1.087 patients will be collected prospectively from approximately 200 sites in Spain. There are planned 6 participating autonomous communities: Madrid, Cataluña, Galicia, Andalucía, Comunidad Valenciana and País Vasco.

#### 9.2.1 Selection of sites:

Cardiologists and non-cardiologist sites regularly prescribing Pradaxa® and VKA for stroke prevention in non-valvular atrial fibrillation according to the respective Summary of Product Characteristics will participate.

Selected sites should include those physicians (e.g. cardiologists, non-cardiologists) and facilities (e.g. specialist offices, hospitals, outpatient care centres etc.) that reflect the clinical practice. These site selection criteria will help to ensure that the patients recruited into that study will represent the patients treated in Spain.

After initiation, every site should include the first consecutive suitable patients where decision for switch to Pradaxa® has been made. The inclusion of the patient in the study is not related with the decision of dabigatran prescription. Dabigatran prescription is based in the Health authorities' recommendations in the positiong

**report of NACOs.** In consecutive sampling, every eligible patient is selected until the required sample size is enrolled. This approach helps to reduce the likelihood of selection bias.

The decision for therapy has to be taken prior and independently of enrolment into the study.

Patients will have to sign informed consent before they can take part in the non-interventional study.

A log of all patients included into the study (i.e. having given informed consent) will be maintained in the ISF at the investigational site irrespective of whether they complete the assessments or not.

#### 9.2.2 Inclusion criteria:

- Written informed consent prior to participation
- Female and male patients  $\geq$ 18 years of age with a diagnosis of non-valvular atrial fibrillation.
- At least 6 months of continuous VKA treatment for stroke prevention prior to baseline assessment.
- Patients switched to Pradaxa® according to Summary of Product Characteristics, therapeutic positioning report from Spanish competent authorities and visa from each autonomous community.
- The inclusion of the patient in the study is not related with the decision of dabigatran prescription. Dabigatran prescription is based in the Health authorities recommendations in the positiong report of NACOs

## 9.2.3 Exclusion criteria:

- Contraindication to the use of Pradaxa® or VKA as described in the Summary of Product Characteristics (SmPC).
- Patients receiving Pradaxa® or VKA for any other condition than stroke prevention in non-valvular atrial fibrillation.
- Current participation in any clinical trial of a drug or device.

## 9.2.4 Removal of patients from the study

Every patient has the right to withdraw consent at any time during the study, without the need for justification and without any impact on the routine therapy.

Boehringer Ingelheim reserves the right to discontinue the study overall or at a particular study site at any time for the following reasons:

- 1. Failure to meet expected enrolment goals overall or at a particular study site.
- 2. Emergence of any efficacy/safety information that could significantly affect continuation of the study, or any other administrative reasons.
- 3. Violation of the protocol, or the contract by a study site or investigator, disturbing the appropriate conduct of the study.

## 9.2.5 Visit schedule

Collection of patient data should be managed during routine practice visits. The timeschedule below can only be a recommendation; if a patient does not visit the site at these time points, data will not be collected (no visits will be conducted solely for study purposes).

Visits cannot be performed by phone as the patient has to complete the self-administered questionnaires.

- 1. At Baseline (at initiation on Pradaxa®)
- 2. 30-45 days after initiation on Pradaxa® (initiation period)
- 3. 150-210 days after initiation on Pradaxa® (continuation period)

Table 9.2: 1 Schedule of Data Collection

| Assessment | Baseline | 30-45 days | 150 –210 days |
|---|---|---|---|
| Inclusion/exclusion criteria | х | | |
| Patient demographics: age, gender | X | | |
| Concomitant diseases | x | | |
| Concomitant therapies | X | X | X |
| HAS- BLED score (to<br>be calculated in the<br>eCRF) | x | | |
| CHA <sub>2</sub> DS <sub>2</sub> -VASc score<br>(to be calculated in the<br>eCRF) | x | | |
| Assessment of duration of previous VKA treatment | х | | |
| Reasons for switch to Pradaxa® | х | | |
| Pradaxa® dosing (110 or 150 mg) and reasons for dose changes | х | х | х |
| Creatinine clearance calc. via Cockcroft-Gault Formula (Creatinine values if available from already existing lab report) to be calculated in eCRF) | х | | |
| ADR, SAE collection | | х | X |
| Reason for Pradaxa® discontinuation | | X | X |

## Boehringer Ingelheim Non-interventional Study Protocol BI Study Number 1160.253


| PACTQ- 2 questionnaire | X | X | X |
|------------------------|---|---|---|
|------------------------|---|---|---|

#### **Baseline visit:**

No data collection for study purposes must be performed unless the patient has consented to participate in the study. Once the patient has signed the informed consent form, the patient is considered to be enrolled in the study and patient details should be recorded on the enrolment log.

The following procedures will be performed at the baseline visit:

- Sign informed consent form
- Review of inclusion and exclusion criteria
- Collection of demographic data: age, gender,
- Collection of current concomitant diseases
- Collection of current concomitant therapies
- Weight will be measured for calculation of creatinine clearance
- Creatinine Clearance: serum creatinine value (if available) to be entered on eCRF, Creatinine Clearance according to Cockcroft-Gault formula to be automatically calculated
- CHA<sub>2</sub>DS<sub>2</sub>-VASc and HAS-BLED score calculation in eCRF
- Duration of previous treatment with VKA to be documented
- Reasons for switch to Pradaxa® to be documented
- Documentation of Pradaxa® dosing
- Patient will be asked to complete the following patient related questionnaires:
  - PACTQ-2
- Treatment with Pradaxa® it was initiated. The inclusion of the patient in the study is not related with the decision of dabigatran prescription. Dabigatran prescription is based in the Health authorities recommendations in the positiong report of NACOs.

#### **Initiation period:**

During a routine practice visit occurring at 30–45 days after initiation of treatment, the following assessments will be documented:

- Current dosing of Pradaxa® and reasons for dose change (if applicable)
- Changes in concomitant therapies
- Collection and reporting of ADR, SAEs (if applicable)
- Reasons for Pradaxa® discontinuation (if applicable)
- Patients will be asked to complete the PACTQ-2 questionnaire

## **Continuation period:**

During a routine practice visit occurring at 150-210 days after initiation of treatment, the following assessments will be documented:

- Current dosing of Pradaxa® and reasons for dose change (if applicable)
- Changes in concomitant therapies
- Collection and reporting of ADR, SAEs (if applicable)
- Reasons for Pradaxa® discontinuation (if applicable)
- Patients will be asked to complete the PACTQ-2 questionnaire

With this visit, the patient's participation in the study will be completed.

## **Description and justification of patient questionnaires:**

## - PACT-Q:

The PACT-Q was developed as a means to investigator patients satisfaction with anticoagulant treatment and treatment convenience in patients with deep venous thrombosis (DVT), pulmonary embolism (PE) or atrial fibrillation (AF). The PACT-Q is a self-administered questionnaire. It can be completed in about ten minutes. No specific training is required to complete this document.

## 9.2.6 Treatments

Patients will be switched from standard care VKA treatment to Pradaxa®

- Pradaxa® 110 mg hard capsules
- Pradaxa® 150 mg hard capsules

Pradaxa® 110 mg and Pradaxa® 150 mg hard capsules contain Dabigatran etexilate (active ingredient: Dabigatran).

Patients will receive daily dose of Pradaxa® according to the Summary of Product characteristics, therapeutic positioning report from Spanish competent authorities and visa from each autonomous community.

The current version of Pradaxa® Summary of Product Characteristics (SmPC) can be found on the EMA Webpage.

The following link is updated with the most recent version of the approved SmPC: <a href="http://ec.europa.eu/health/documents/community-register/html/h442.htm">http://ec.europa.eu/health/documents/community-register/html/h442.htm</a>

#### 9.2.7 Concomitant medications and restrictions

All concomitant medications are prescribed based on the underlying medical condition and upon the discretion of the treating physician. No treatment will be withheld from the patients. Any prescription is in the responsibility of the treating physician.

## 9.2.8 Representativeness of the study population:

Inclusion and exclusion criteria have been limited to the respective SmPCs of Pradaxa®. Therefore the patient population recruited in this non-interventional study can be seen as representative for patients receiving VKA therapy and subsequent initiation of treatment with Pradaxa® for stroke prevention in non-valvular atrial fibrillation.

## 9.4 VARIABLES

## 9.4.1 Primary objective:

<u>Outcome 1:</u> Mean PACT-Q2 scores at second and last assessment compared to baseline assessment.

**Outcome 2:** Mean PACT-Q2 score at last assessment compared to second assessment.

#### 9.4.2 For Secondary objectives

Outcome 1: Characterization of patients according to

- Age
- Gender
- CHA<sub>2</sub>DS<sub>2</sub>-VASc score (R10-5332)
- HAS-BLED score (R10-6394)
- Kidney function (creatinine clearance)
- Stroke and/or bleeding related risk factors in medical history and at baseline
- Concomitant diseases
- Concomitant therapies
- Dosing of Pradaxa®
- Duration of previous VKA treatment

#### 9.5 DATA SOURCES

Data will be newly collected. Patients will be asked to complete the respective questionnaires during their routine visits. Patient demographic data, concomitant diseases and concomitant therapies will be completed based on the physician's records. Information on Pradaxa® and/or VKA dosing will be collected from physician's records. Creatinine clearance for assessment of kidney function will be calculated within the eCRF, by entering Creatinine values (from existing lab reports, if available), and weight to be measured by the physician.

## 9.6 STUDY SIZE

It is planned that a total of 1.807 patients from Spain will be recruited for the study. The planned total sample size is jointly determined by the following sample size calculations and additional non-statistical considerations, including feasibility assessments for each participating autonomous community.

Baseline characteristics and other pre-specified attributes of the patient population will be described by estimates and confidence intervals for all patients

Categorical attributes will be estimated with the precision (i.e. width of descriptive 95% confidence interval) described in Table 9.6:1, according to sample size and prevalence of the attribute.

Table 9.6: 1 Width of 95% confidence interval\* by sample size and prevalence of attribute

| Prevalence of attribute | | Sample size (total or subgroup) | | | | | |
|---|---|---|---|---|---|---|---|
| | | 100 | 200 | 500 | 800 | 1.000 | 1.087 |
| 10% | Expected n | 10 | 20 | 50 | 80 | 100 | 109 |
| | 95% CI width | 12.72 | 8.80 | 5.46 | 4.28 | 3.82 | 3.66 |
| 20% | Expected n | 20 | 40 | 100 | 160 | 200 | 218 |
| | 95% CI width | 16.51 | 11.53 | 7.20 | 5.66 | 5.05 | 4.84 |
| 30% | Expected n | 30 | 60 | 150 | 240 | 300 | 327 |
| | 95% CI width | 18.74 | 13.13 | 8.21 | 6.47 | 5.77 | 5.53 |
| 40% | Expected n | 40 | 80 | 200 | 320 | 400 | 435 |
| | 95% CI width | 19.95 | 13.99 | 8.77 | 6.90 | 6.17 | 5.91 |
| 50% | Expected n | 50 | 100 | 250 | 400 | 500 | 544 |
| | 95% CI width | 20.34 | 14.26 | 8.94 | 7.04 | 6.29 | 6.03 |

<sup>\*</sup> Calculations are based on the Clopper-Pearson method.

For example, for a population attribute with a prevalence of 20%, a sample size of 1.087 patients allows this proportion to be estimated with a precision of 4.84% (i.e. width of 95% CI). As another example, for a population attribute with a prevalence of 30%, a specific sample size for a group of 500 patients allows this proportion to be estimated with a precision of 8.21%.

Due to the limited number of publications on PACT-Q (studies to be referenced: (R15-1314, R15-1316) (R15-1359) and the lack of information regarding the clinical meaning of PACT-Q scale changes, sample sizes are estimated with the use of standardized mean differences. In the context of this study, they represent the mean differences in PACT-Q scores between two time points divided by the corresponding standard deviations. In general, a standardized effect size of 0.2 is considered a small change, 0.5 a moderate change, and 0.8 a large change.

Assuming a 2-sided alpha of 0.05 and a 20% loss to follow-up, a sample size of 1.087 patients will provide 90% power to detect a standardized mean difference of 0.11 for the primary endpoint of PACT-Q2 scores between the last and baseline assessments.

Based on results reported in the PREFER in AF (R15-1312) registry study, a reasonable expected standard deviation for the mean convenience and treatment satisfaction scores is 16. Using this estimate, Table 9.6:2 shows the conversion of various standardized

## Boehringer Ingelheim Non-interventional Study Protocol BI Study Number 1160.253


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

mean differences to actual mean differences in the convenience and treatment satisfaction scores.

Table 9.2: 2 Conversion of standardized mean difference to actual mean difference in the convenience and treatment satisfaction scores (assuming a standard deviation of 16)

| Standardized mean difference | Actual mean difference in the convenience and treatment satisfaction scores |
|---|---|
| 0.1 | 1.6 |
| 0.2 | 3.2 |
| 0.3 | 4.8 |
| 0.4 | 6.4 |
| 0.5 | 8.0 |

#### 9.7 DATA MANAGEMENT

A data management plan (DMP) will be created to describe all functions, processes, and specifications for data collection, cleaning and validation. The electronic CRFs (eCRFs) will include programmable edits to obtain immediate feedback if data are missing, out of range, illogical or potentially erroneous. These rules may encompass simple checks such as range validation or presence/absence of data, or concurrent manual data review may be performed based on parameters dictated by the DMP. Ad hoc queries to the sites may be generated and followed up for resolution. A source data quality audit may be initiated to ensure that the data in the database is accurate.

The database will be housed in a physically and logically secure computer system maintained in accordance with a written security policy. The system will meet the standards of the International Committee on Harmonization guideline E6R1 regarding electronic study data handling. Patient confidentiality will be strictly maintained.

## 9.8 DATA ANALYSIS

#### 9.8.1 STUDY DESIGN

In this non-interventional study, cross-sectional data at study baseline and longitudinal follow-up data over 6 months will be collected for non-valvular AF patients with a VKA therapy and subsequent initiation of Pradaxa®.

Baseline data will be described using a cross-sectional approach. Data from the longitudinal follow-up will be summarized descriptively. Mean difference in PACT-Q2 scores between assessment time points will be assessed. Due to the nature of this non-interventional study, there is no (confirmatory) hypothesis testing foreseen in a strict statistical sense. Analyses are descriptive in nature and confidence intervals and p-values from statistical models are used for exploratory purposes. No adjustments for multiple testing are made in the evaluation of statistical significance. Consequently, significant differences may be observed by chance alone and p-values should be interpreted as exploratory and with caution.

#### 9.8.2 PLANNED ANALYSES

Analyses will be performed by Boehringer Ingelheim's designees. The main analysis population will consist of all eligible patients (i.e. all patients fulfilling all inclusion criteria and no exclusion criteria).

Summary statistics for continuous variables will include the N, mean, standard deviation, minimum, Q1 (lower quartile), median, Q2 (upper quartile), and maximum value; tabulations of categorical variables will present all possible categories and will display the number of observations per category as well as percentages. Estimates will be presented with 95% confidence intervals for the variables of interest.

Additional details of the planned analysis will be provided in the statistical and epidemiological analysis plan (SEAP).

## 9.8.2.1 Main Analyses

Patient demographics and disease characteristics at baseline as described in section 8.3.2 will be summarized descriptively for all eligible patients in the study. This analysis may be repeated by additional relevant factors that will be specified in the SEAP. If deemed appropriate, continuous and categorical variables may be compared between groups using t-tests (or non-parametric tests) and chi-square tests, respectively.

The primary outcome of the mean difference in PACT-Q2 scores between the last and baseline assessment will be analyzed using a paired t-test (or the non-parametric Wilcoxon test for non normal distributed data). The primary analyses will be based on the actual anticoagulation treatment the patients receive (i.e. "as treated" analysis). A patient is considered to have permanently discontinued initial anticoagulation treatment if other relevant anticoagulation treatment is initiated or otherwise dependent on the duration of treatment interruption (details will be provided in the SEAP). Patients who have permanently discontinued initial anticoagulation treatment at the time of an assessment will be excluded from all analyses where data from that assessment is included.

## 9.8.2.2 Further Analyses

Mean differences in PACT-Q2 between other assessment time points will be analyzed using the same statistical procedure as described for the primary endpoint.

## 9.8.2.3 Safety Analyses

Safety analyses will include all enrolled patients with an actual follow-up. Statistical analysis and reporting of AEs will be descriptive in nature, will be based on BI standards, and will focus on adverse drug reactions (i.e. AEs related to anticoagulation treatment). No hypothesis testing is planned.

Occurrences of AEs will be analyzed relative to the number of patients treated as well as observed person-years (i.e. time at risk). Safety analysis will be based on the concept of treatment emergent AEs. Patients will be analyzed according to the anticoagulation treatment received at the time of the event. If no concurrent anticoagulation treatment is administered, then events occurring within a washout period of 6 days after discontinuation of anticoagulation treatment will be assigned to the last treatment given. This washout period will also be included as time at risk for derivation of total person-years. AEs that deteriorate under treatment will also be considered as "treatment emergent". AEs occurring prior to first intake of anticoagulation treatment prescribed at baseline, during periods without any anticoagulation treatment (excluding washout periods), or after the end of the 6 month follow-up (excluding washout periods) will not be considered treatment emergent events and will not be included in the summary tables.

The following parameters will be included in the safety analyses:

- Adverse drug reactions
- Adverse drug reactions leading to discontinuation of anticoagulation treatment
- Serious adverse drug reactions
- Deaths
- SAEs

## 9.8.2.4 Schedule of Planned Analyses

All planned analyses as specified in Section 9.8.2.1 to 9.8.2.3 will be performed once the data collection is completed, the data sets are cleaned, and the database is locked. One final report will be prepared at the completion of the study.

#### 9.8.3 HANDLING OF MISSING DATA

Every reasonable attempt will be undertaken to ensure completeness of data collection. Imputation will be permitted, if deemed appropriate and on a case-by-case basis, depending on the extent and distribution of missing values, and will be described in the SEAP.

The percentage of and reason for loss to follow-up will be summarized overall, and by other relevant factors if deemed appropriate. In addition, if the proportion of patients with loss to follow-up is substantial enough (e.g.  $\geq 10\%$ ) to warrant further investigation, baseline characteristics will be described for patients who were lost to follow-up in comparison to patients who have completed follow-up.

## 9.9 QUALITY CONTROL

The following processes will be implemented to ensure data completeness and data quality:

## **Data Edit Checks:**

The electronic CRF (eCRF) will include programmable edit checks to obtain feedback if data is missing, out of range, illogical or potentially erroneous.

These checks will be performed once data is entered into the eCRF.

Thus the data entered in to the eCRF will be validated within the system and the physician will receive alerts for missing or inconsistent data. In case any changes of already entered data will be required, an audit trail will be available.

#### **Medical monitoring:**

A review of applicable entered eCRF data will be performed to verify patient eligibility to ensure that the analysed patient population corresponds to the protocol–described population.

In addition, the CRO will also review eCRFs/completed patient related questionnaires for verification that no non reported safety event is present.

## Source data verification:

No regular source data verification is planned in this non-interventional study. However, in case of issues (i.e. high amount of missing data, data discrepancies, protocol violations etc) detected at a site with the measures described above, a for-cause onsite visit can be planned to perform a sample check of source data.

#### 9.10 LIMITATIONS OF THE RESEARCH METHODS

## Boehringer Ingelheim Non-interventional Study Protocol BI Study Number 1160.253

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Consecutive enrolment will be employed to ensure that specific types of patients are not selected by site staff to participate.

VKA has been the mainstay of SPAF for many years. It is widely available, affordable but does require regular INR monitoring. Pradaxa® is more expensive, may or may not be reimbursed but doesn't require the continual INR monitoring. There are a number of different types of bias that could influence the data collection and analysis from the study such as selection bias or recall bias.

The study is designed to collect new data. The entry criteria are non-restrictive which will permit the enrolment of a broad patient population. The choice of treatment is at the discretion of the investigator. Therefore the data collected in this study should reflect the real world treatment patterns and patient characteristics.

#### **Selection bias:**

Selection bias could occur at both the site level and the patient level. If sites where Pradaxa® is used frequently differ systematically with respect to patient or the routine procedures from sites that use Pradaxa® less frequently, the between site difference could lead to non-comparability between the patients. To minimize the site level selection bias, the goal is to have participating centres that have access to all available treatment options for SPAF that are approved for use in that country.

Selection bias at the patient level could occur if sites preferentially enroll specific patients into the study. To minimize selection bias at the patient level, consecutive enrolment is performed.

#### Loss to follow-up:

All efforts will be made to minimize loss to follow-up in patients who are enrolled. Patients who are lost to follow-up will be characterized and compared to the remaining patients and the reason and time point of lost to follow-up will be evaluated.

#### Recall bias:

Recall bias refers to the phenomenon when the outcomes of treatment (either good or bad) may colour the patient's recollection of events prior to or during the treatment. To minimize recall bias, patient reported outcomes will be assessed using validated scales within a limited period of time to minimize recall bias.

#### **Confounding:**

Confounding occurs when an observed association is due to three factors: the exposure, the outcome of interest and a third factor which is independently associated with both the outcome of interest and the exposure. Statistical techniques, such as adjustment for covariates may be used to correct for identified confounders. However unidentified confounders cannot be controlled for using statistical analysis.

#### 9.11 OTHER ASPECTS

#### 9.11.1 INFORMED CONSENT, DATA PROTECTION, STUDY RECORDS

The study will be carried out in compliance with the protocol, the principles laid down in the Declaration of Helsinki, and relevant BI Standard Operating Procedures (SOPs). Standard medical care (prophylactic, diagnostic and therapeutic procedures) remains in the responsibility of the treating physician of the patient.

The investigator should inform the sponsor immediately of any urgent safety measures taken to protect the study subjects against any immediate hazard, and also of any serious breaches of the protocol.

The rights of the investigator and of the sponsor with regard to publication of the results of this study are described in the investigator contract. As a general rule, no study results should be published prior to finalization of the Study Report.

# 9.11.1.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT

This study will be initiated only after all required legal documentation has been reviewed and approved by the respective Independent Ethics Committee (IEC) and competent authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments.

Prior to patient participation in the study, written informed consent must be obtained from each patient (or the patient's legally accepted representative) according to the regulatory and legal requirements of Spain. Each signature must be personally dated by each signatory and the informed consent and any additional patient-information form retained by the investigator as part of the study records. A signed copy of the informed consent and any additional patient information must be given to each patient or the patient's legally accepted representative.

The patient must be informed that his/her personal study-related data will be used by Boehringer Ingelheim in accordance with the local data protection law. The level of disclosure must also be explained to the patient.

The patient must be informed that his / her medical records may be examined by authorized monitors (CML/CRA) or Clinical Quality Assurance auditors appointed by Boehringer Ingelheim, by appropriate IEC members, and by inspectors from regulatory authorities.

## 9.11.1.2 DATA QUALITY ASSURANCE

A quality assurance audit/inspection of this study may be conducted by the sponsor or sponsor's designees or by IECs or by regulatory authorities. The quality assurance

## Boehringer Ingelheim Non-interventional Study Protocol BI Study Number 1160.253

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

auditor will have access to all medical records, the investigator's study-related files and correspondence, and the informed consent documentation of this study.

## 9.11.1.3 RECORDS

Case Report Forms (CRFs) for individual patients will be provided by the sponsor via remote data capture. All of the clinical data and site/investigator characteristics will be captured via a web-based EDC system. The site staff will enter and edit the data via a secure network, with secure access features (username, password and secure identification – an electronic password system). A complete electronic audit trail will be maintained. The Investigator will approve the data using an electronic signature that is 21 CFR Part 11 compliant.

Patients must not be identified on the eCRF by name. Appropriately coded identification (i.e. Patient numbers) must be used. The Investigator must make a separate confidential record of these details (Patient enrollment log) to permit the identification of all patients enrolled in the study in case follow-up is required. Any supporting documentation must be redacted of any patient identifying information and the patient ID number must be clearly written on the documents.

#### 9 11 1 3 1 Source documents

Source documents provide evidence for the existence of the patient and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.

Data entered in the eCRFs that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study; also current medical records must be available.

For eCRFs all data must be derived from source documents.

#### 9.11.1.3.2 Direct access to source data and documents

The investigator / institution will permit study-related monitoring, audits, IEC review and regulatory inspection, providing direct access to all related source data / documents. eCRFs and all source documents, including progress notes and copies of laboratory and medical test results must be available at all times for review by the sponsor's clinical study monitor, auditor and inspection by health authorities (e.g. AEMPS). The Clinical Research Associate (CRA) and auditor may review all eCRFs, and written informed consents. The accuracy of the data will be verified by reviewing the documents described in Section 8.10.1.3.1.

#### 9.11.1.4 STATEMENT OF CONFIDENTIALITY

Individual patient medical information obtained as a result of this study is considered confidential and disclosure to third parties is prohibited with the exceptions noted below. Patient confidentiality will be ensured by using patient identification code numbers.

## Boehringer Ingelheim Non-interventional Study Protocol BI Study Number 1160.253


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Treatment data may be given to the patient's personal physician or to other appropriate medical personnel responsible for the patient's welfare. Data generated as a result of the study need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IEC and the regulatory authorities.

## 9.11.1.5 COMPLETION OF STUDY

The EC/competent authority needs to be notified about the end of the study (last patient out), or early termination of the study.

# 10. PROTECTION OF HUMAN SUBJECTS

Please refer to section 8.10.1

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

#### 11.1 DEFINITIONS OF ADVERSE EVENTS

#### Adverse event:

An adverse event (AE) is defined as any untoward medical occurrence, including an exacerbation of a pre-existing condition, in a patient in a clinical investigation who received a pharmaceutical product. The event does not necessarily have to have a causal relationship with this treatment.

## Serious adverse event:

A serious adverse event (SAE) is defined as any AE which results in death, is immediately life-threatening, results in persistent or significant disability / incapacity, requires or prolongs patient hospitalization, is a congenital anomaly / birth defect, or is to be deemed serious for any other reason if it is an important medical event when based upon appropriate medical judgment which may jeopardize the patient and may require medical or surgical intervention to prevent one of the other outcomes listed in the above definitions.

#### Intensity of adverse event:

The intensity of the AE should be judged based on the following:

Mild: Awareness of sign(s) or symptom(s) which is/are easily tolerated Moderate: Enough discomfort to cause interference with usual activity

Severe: Incapacitating or causing inability to work or to perform usual activities

## Causal relationship of adverse event:

Medical judgment should be used to determine the relationship, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or rechallenge, confounding factors such as concomitant medication, concomitant diseases and relevant history. Assessment of causal relationship should be recorded in the case report forms.

Yes: There is a reasonable causal relationship between the investigational product administered and the AE.

No: There is no reasonable causal relationship between the investigational product administered and the AE.

Worsening of the underlying disease or other pre-existing conditions.

Worsening of the underlying disease or of other pre-existing conditions will be recorded as an

(S)AE in the (e)CRF.

## Boehringer Ingelheim Non-interventional Study Protocol BI Study Number 1160.253

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Changes in vital signs, ECG, physical examination, and laboratory test results.

Changes in vital signs, ECG, physical examination and laboratory test results will be recorded as an (S)AE in the (e)CRF, if they are judged clinically relevant by the investigator.

#### 11.2 ADVERSE EVENT AND SERIOUS ADVERSE EVENT REPORTING

All adverse events, serious and non-serious, occurring during the course of the clinical trial (i.e., from signing the informed consent onwards through the observational phase) will be collected, documented and reported to the sponsor by the investigator on the appropriate eCRFs / SAE reporting forms. Reporting will be done according to the specific definitions and instructions detailed in the 'Adverse Event Reporting' section of the Investigator Site File.

For each adverse event, the investigator will provide the onset date, end date, intensity, treatment required, outcome, seriousness, and action taken with the investigational drug. The investigator will determine the relationship of the investigational drug to all AEs as defined in Section 10.1

The investigator also has the responsibility to report AEs occurring in 30 days after a patient completes the trial. Any AEs reported to the sponsor during this phase must be documented in the safety database.

The investigator must report the following events via fax using the SAE form within the following timelines:

- Fatal AEs, life threatening ADRs (plus non-serious AEs that are part of a serious ICSR): day 0,
- Serious ADRs (plus Non-serious AEs that are part of a serious ICSR): day 1
- Non-serious ADRs /DEDP: day 7, aggregated or as single reports.

The Investigator must carefully assess whether AE constitutes an ADR. The term AE includes Drug exposure during pregnancy (DEDP). The investigator would report an AE and would indicate whether administration of study medication was correct and if not indicate the appropriate, e.g. overdose, abuse, misuse, medication error, occupational exposure, lack of effect, unexpected benefit.

The SAE form is to be forwarded to the defined unique entry point (contact details will be provided in the Investigator Site File). It also applies if new information to existing SAEs or protocol-specified significant events becomes available.

All other Adverse Events must be reported on the (e)CRFs within 2 weeks to the Sponsor. CRFs have to be forwarded to the defined database site (contact details will be provided in the Investigator Site File).

#### Pregnancy:

The investigator must report any drug exposure during pregnancy to the sponsor to the defined unique entry point for SAE forms (contact details will be provided in the Investigator Site File). The outcome of the pregnancy associated with the drug exposure during pregnancy must be followed up. In the absence of an (S) AE, only the Pregnancy Monitoring Form and not the SAE form is to be completed. The ISF will contain the Pregnancy Monitoring Form (Part A and Part B).

#### 11.3 TIME WINDOWS

To fulfil the regulatory requirements for expedited safety reporting, the sponsor evaluates whether a particular adverse event is "listed", i.e. is a known side effect of the drug or not. Therefore a unique reference document for the evaluation of listedness needs to be provided. For Pradaxa® this is EU SmPC for Pradaxa®; the current versions of these reference documents are available on the EMA homepage: <a href="http://ec.europa.eu/health/documents/community-register/html/h442.htm">http://ec.europa.eu/health/documents/community-register/html/h442.htm</a>
# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

Results of this non-interventional study will be disclosed on external websites according to BI SOP.

In addition, a study specific publication plan will be developed to describe planned publications for overall study results.

#### 13. REFERENCES

#### 13.1 PUBLISHED REFERENCES

- P13-05668 Monz BU, Connolly SJ, Korhonen M, Noack H, Pooley J Assessing the impact of dabigatran and warfarin on health-related quality of life: results from an RE-LY sub-study. Int J Cardiol 168 (3), 2540 2547 (2013).
- R10-5332 Lip GYH, Nieuwlaat R, Pisters R, Lane DA, Crijns HJGM Refining clinical risk stratification for predicting stroke and thromboembolism in atrial fibrillation using a novel risk factor-based approach: the Euro Heart Survey on Atrial Fibrillation. Chest 137 (2), 263 272 (2010).
- R10-6394 Pisters R, Lane DA, Nieuwlaat R, Vos CB de, Crijns HJGM, Lip GYH A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest 138 (5), 1093 1100 (2010).
- R15-1312 Caterina R de, Brueggenjuergen B, Darius H, Heuzey JY le, Renda G, Schilling RJ, Schmitt J, Zamorano JL, Kirchhof P Quality of life and patient satisfaction data in atrial fibrillation patients stably treated with a VKA vs patients switched from a VKA to NOAC. The PREFER in AF registry. ESC 2014, 36th Cong of the European Society of Cardiology (ESC), Barcelona, 30 Aug 3 Sep 2014 (Poster)
- R15-1314 Prins MH, Guillemin I, Gilet H, Gabriel S, Essers B, Raskob G, Kahn SR Scoring and psychometric validation of the Perception of Anticoagulant Treatment Questionnaire (PACT-Q).

  Health Qual Life Outcomes 7, 30 (2009)
- R15-1316 Prins MH, Marrel A, Carita P, Anerson D, Bousser MG, Crijns H, Consoli S, Arnould B Multinational development of a questionnaire assessing patient satisfaction with anticoagulant treatment: the 'Perception of Anticoagulant Treatment Questionnaire' (PACT-Q). Health Qual Life Outcomes 7, 9 (2009)
- R15-1350 Oemar M, Janssen B EQ-5D-5L user guide: basic information on how to use the EQ-5D-5L instrument (version 2.0, October 2013). http://www.euroqol.org/fileadmin/user\_upload/Documenten/PDF/Folders\_Fly ers/UserG uide\_EQ-5D-5L\_v2.0\_October\_2013.pdf (access date: 24 March 2015);Rotterdam: EuroQol Group (2013)
- R15-1359 Heidorn K, Haenschke J, Lindner T, Mittelmeier W, Skripitz R Health economic analysis of thromboprophylaxis with rivaroxaban and certoparin-sodium in patients after total hip or knee replacement. Int J Orthop 1 (1), 15 18 (2014)

#### 13.2 UNPUBLISHED REFERENCES

None.

#### ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

# PACT-Q2 (Perception AntiCoagulant Treatment Questionnaire)

- The purpose of this questionnaire is to understand your expectations and to assess your satisfaction with your anticoagulant treatment (treatment that stops the blood from clotting).
- Throughout the questionnaire, the term "taking" refers to how you take your anticoagulant treatment (either by pill or injection).
- Please read each question carefully, answering as openly as you can and without help from anyone. There are no wrong answers.
- All of the information you provide will be kept confidential.
  - This questionnaire will take about **10 minutes** to complete.

#### Convenience

Please answer the following questions to help us understand how convenient it is to take your treatment.

#### Please check one box per line.

B1 - How difficult is it to take your anticoagulant treatment (i.e., pills or injections, number of pills or injections, frequency of intake ...)?

| $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
|-------------|-------------|-------------|-------------|-------------|
| Not at all | A little | Moderately | A lot | Extremely |

B2 - How bothered are you by taking your anticoagulant treatment?

| | $\square_2$ | | $\square_3$ | | $\square_4$ | | |
|------------|-------------|---|-------------|---|-------------|---|-----------|
| Not at all | A little | M | oderately | U | Alot | 7 | Extremely |

B3 Some anticoagulant treatments may need dose adjustments; how difficult is this for you?

| $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
|-------------|-------------|-------------|-------------|-------------|
| Not at all | A little | Moderately | A lot | Extremely |

B4 - Certain medications CANNOT be taken with anticoagulant treatments; how difficult is this for you?

| $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
|-------------|-------------|-------------|-------------|-------------|
| Not at all | A little | Moderately | A lot | Extremely |

| $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | |
|---|---|---|---|---|
| Not at all | A little | Moderately | A lot | Extremely |
| ow difficult is ome? | it for you to tal | ke your anticoagul | ant treatment | when you are av |
| $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | |
| Not at all | A little | Moderately | A lot | Extremely |
| Not at all | th nurses, doctor $\square_2$ A little | rs or labs)? \$\Bigsize \Pi_3\$ Moderately | A lot | Extremely |
| Not at all ow bothered eatment? | A little | □ <sub>3</sub> Moderately e medical follow- | A lot | Extremely with your anti- |
| Not at all ow bothered teatment? $\Box_1$ | A little are you by the $\Box_2$ | □ <sub>3</sub> Moderately e medical follow- | A lot -up required □4 | Extremely with your antic $\square_5$ |
| Not at all low bothered reatment? | A little | □ <sub>3</sub> Moderately e medical follow- | A lot | Extremely with your anti- |
| Not at all Not at all low bothered reatment? □ 1 Not at all | A little A little $\Box_2$ A little $\Delta_2$ A little | □ <sub>3</sub> Moderately e medical follow- | A lot -up required □4 A lot | Extremely with your antic |
| Not at all Not at all low bothered reatment? In the second of the sec | A little A little $\Box_2$ A little $\Delta_2$ A little | Moderately e medical follow- Moderately Moderately | A lot -up required □4 A lot | Extremely with your antic |

B10 - Do you feel more dependent on others (i.e partner, family, nurse...) because of your anticoagulant treatment?

| $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
|-------------|-------------|-------------|-------------|-------------|
| Not at all | A little | Moderately | A lot | Extremely |

B11 - How worried are you about having to interrupt or stop your anticoagulant treatment?

| $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
|-------------|-------------|-------------|-------------|-------------|
| Not at all | A little | Moderately | A lot | Extremely |

# REVIEW COPY Do not use without permission

#### **Burden of Disease and Treatment**

Please answer the following questions to help us understand how your disease and its treatment affect you.

#### Please check one box per line.

C1 - Because of potential side effects (i.e., minor bruises, bleeding...), do you limit your usual activities (i.e., work, leisure, social, or physical activities...)?

| | $\square_2$ | $\square_3$ | | | 5 | |
|------------|-------------|-------------|-------|--------|------|-----|
| Not at all | A little | Moderately | A lot | Extren | nely | 551 |

C2 - How much physical discomfort do you have due to bruises or pain?



## **Anticoagulant Treatment Satisfaction**

Please answer the following questions to help us understand how satisfied you are with your treatment.

#### Please check one box per line.

D1 - How reassured do you feel by your anticoagulant treatment?

| | $\square_2$ | $\square_3$ | $\Box_4$ | $\square_5$ |
|------------|-------------|-------------|----------|-------------|
| Not at all | A little | Somewhat | Very | Completely |

D2 - Do you feel that your anticoagulant treatment has decreased your symptoms (i.e., leg pain or swelling, palpitations, shortness of breath, or chest pain...)?

| | $\square_1$ | U | | $\square_2$ | | $\square_3$ | | $\square_4$ | $\square_5$ |
|---|---|---|---|---|---|---|---|---|---|
| No | ot at a | 11 | A | little | ; | Moderately | I | A lot | Completely |

D3 - How did your experience with side effects such as minor bruises or bleeding (i.e., while shaving, cooking, after small cuts...) compare to what you expected?

| $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
|---|---|---|---|---|
| It is much<br>worse than<br>what I<br>expected | It is worse<br>than what I<br>expected | It is exactly what I expected | It is better<br>than what I<br>expected | It is much<br>better than<br>what I<br>expected |

| D4 - | Regarding the follow-up of your disease and anticoagulant treatment, how satisfied are | e |
|---|---|---|
| | you with your level of independence? | |

| $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
|---|---|---|---|---|
| Extremely dissatisfied | Dissatisfied | Neither<br>satisfied nor<br>dissatisfied | Satisfied | Extremely satisfied |

D5 - How satisfied are you with the methods (i.e., appointments with nurses, doctors, labs...) used to ensure the follow-up of your disease and anticoagulant treatment?

| | $\square_2$ | $\square_3$ | $\square_4$ | |
|---|---|---|---|---|
| Extremely dissatisfied | Dissatisfied | Neither<br>satisfied nor<br>dissatisfied | Satisfied | Extremely satisfied |

D6 - How satisfied are you with the form of your anticoagulant treatment (oral pill / injection)?

| $\square_1$ | $\square_2$ | | $\square_4$ | $\square_5$ |
|---|---|---|---|---|
| Extremely dissatisfied | Dissatisfied | Neither<br>satisfied nor<br>dissatisfied | Satisfied | Extremely satisfied |

D7 - **Overall**, how satisfied are you with your anticoagulant treatment?

| | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
|---|---|---|---|---|
| Extremely dissatisfied | Dissatisfied | Neither<br>satisfied nor<br>dissatisfied | Satisfied | Extremely satisfied |

Please make sure you answered all questions.

Thank you for your time.

#### ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

Not applicable for Non interventional studies.

#### **ANNEX 3. ADDITIONAL INFORMATION**

Criteria and general recommendations for the novel oral anticoagulant use for the stroke and systemic embolism prevention in patients with non-valvular atrial fibrillation





# INFORME DE POSICIONAMIENTO TERAPÉUTICO UT/V4/23122013

## Criterios y recomendaciones generales para el uso de nuevos anticoagulantes orales (NACO) en la prevención del ictus y la embolia sistémica en pacientes con fibrilación auricular no valvular

#### Fecha de publicación 23 de diciembre de 2013

La fibrilación auricular (FA) es la arritmia cardiaca crónica más frecuente y se calcula que afecta a un 1-2% de la población [1,2]. Su prevalencia se incrementa con la edad, de modo que se estima que la padece un 8,5% de la población española mayor de 60 años [3].

La FA confiere a los pacientes que la padecen un riesgo de ictus y embolia sistémica superior en 5 veces al de la población general. Se estima que 1 de cada 5 ictus isquémicos están asociados a la presencia de FA. El tratamiento de la FA comprende dos estrategias complementarias. La primera de ellas tiene como objeto recuperar y mantener el ritmo sinusal (control del ritmo) mediante cardioversión eléctrica o farmacológica, que a menudo es seguida de tratamiento antiarrítmico de mantenimiento (FA paroxística recurrente o FA persistente). En segundo lugar, en fases más evolucionadas o situaciones donde el control del ritmo no es una opción posible o se ha desestimado (FA permanente o crónica), la terapéutica se dirige al control de la frecuencia cardiaca, minimizando así la repercusión clínica de la FA. En paralelo, dado que la complicación más importante de la FA por su frecuencia e impacto en la mortalidad prematura y en la discapacidad es el ictus, el tratamiento antitrombótico debe acompañar a ambas estrategias. En presencia de riesgo embólico (ej.: CHADS<sub>2</sub> ≥ 2 puntos) la anticoagulación oral está plenamente indicada, salvo contraindicación formal.

Los antagonistas de la vitamina K (AVK) [acenocumarol (Sintrom®) y warfarina (Aldocumar®)] han sido durante décadas la única opción disponible para la terapia anticoagulante oral (TAO) en la prevención de las complicaciones tromboembólicas de la FA. Tradicionalmente, en pacientes con alguna contraindicación o riesgo especial asociado al uso de los AVK, la alternativa ha sido el tratamiento con antiagregantes plaquetarios [1]. El uso de AVK requiere monitorización del tiempo de protrombina (TP), habitualmente expresado como cociente internacional normalizado (INR). Este y otros factores, tales como el riesgo potencial elevado (a veces sobre-percibido) de interacciones y hemorragias graves, han llevado tradicionalmente a la infrautilización de los AVK en pacientes con FA, si bien el número de pacientes tratados ha ido creciendo considerablemente con el tiempo.

En los últimos años se han desarrollado nuevos medicamentos anticoagulantes, tales como el inhibidor directo de la trombina dabigatrán etexilato (Pradaxa®) [4,5], y los inhibidores directos del factor X activado rivaroxabán (Xarelto®) [6,7] y apixabán (Eliquis®) [8,9], que han demostrado un beneficio-riesgo favorable en diversas condiciones clínicas en las que está indicada la anticoagulación. La utilización de los nuevos anticoagulantes orales (NACO) se asocia con beneficios e inconvenientes respecto del uso de AVK que han sido ya materia de amplia discusión en las evaluaciones de las agencias reguladoras. Dicha evaluación se

confirmará además en los próximos años, con la publicación de resultados de nuevos ensayos clínicos para nuevas condiciones de uso y la experiencia adquirida poscomercialización. Todo ello contribuirá a delimitar de forma más sólida el posicionamiento de estos nuevos medicamentos en la terapéutica.

En el momento actual, surge la necesidad de establecer unas recomendaciones de uso para los NACO, identificando aquellos pacientes en los que las ventajas de estos nuevos tratamientos sean mayores y asegurando que el incremento del número de pacientes tratados se produce de una forma prudente y acompasada con el conocimiento científico sobre estos medicamentos. Asimismo, debe tenerse en cuenta el impacto presupuestario de la sustitución de los AVK por los NACO, que aconseja disponer de un análisis que identifique los grupos de pacientes prioritarios para estos nuevos tratamientos y permita así establecer una estrategia racional para su uso en el Sistema Nacional de Salud (SNS) en las indicaciones autorizadas.

Algunas Comunidades Autónomas han realizado ya algún ejercicio de esta índole para dabigatrán [10-19] y se impone ahora un esfuerzo más global que aglutine los trabajos ya realizados e incluya los tres nuevos anticoagulantes, estableciendo criterios de utilización comunes para todo el SNS, teniendo en cuenta que los AVK siguen siendo la piedra angular en el manejo de estos pacientes. Las recomendaciones del presente informe de posicionamiento terapéutico están basadas en la evidencia disponible. En aquellas situaciones clínicas que involucran pacientes complejos para los que no se dispone ni se prevé se disponga de evidencia sobre el riesgo-beneficio de los NACO obtenida de estudios prospectivos aleatorizados (sección 4.2.1.) las recomendaciones están basadas en la evidencia indirecta disponible y en el consenso del grupo multidisciplinar.

#### 1. EVIDENCIA DE EFICACIA Y SEGURIDAD DE LA ANTICOAGULACIÓN ORAL EN LA PREVENCION DEL ICTUS Y EMBOLIA SISTÉMICA EN PACIENTES CON FIBRILACIÓN AURICULAR Y FACTORES DE RIESGO TROMBOEMBÓLICO ADICIONALES

En pacientes con FA auricular no valvular, los AVK reducen el riesgo de ictus en un 64% en comparación con placebo [20] y, asociados a un seguimiento adecuado, presentan una relación beneficio/riesgo favorable, considerándose coste-efectivos [21]. Los NACO fueron inicialmente aprobados por las agencias reguladoras europeas para la prevención del tromboembolismo venoso (TEV) en pacientes sometidos a cirugía electiva de reemplazo de cadera o rodilla. Con posterioridad, estos medicamentos han sido desarrollados prevención de para la complicaciones tromboembólicas en pacientes con FA y en otras indicaciones (ej.: tratamiento del TEV y síndrome coronario agudo).

Tanto dabigatrán como rivaroxabán y apixabán han sido autorizados en la indicación de prevención del ictus y embolia sistémica en pacientes con FA no valvular (Tabla 1).





| | Pradaxa (dabigatrán) | Xarelto (rivaroxabán) | Eliquis (apixabán) |
|---|---|---|---|
| Indicación | Prevención del ictus y de la embolia sistémica en pacientes adultos con fibrilación auricular no valvular, con uno o más factores de riesgo tales como: Ictus, ataque isquémico transitorio previos Insuficiencia cardíaca ≥ Clase 2 escala New York Heart Association (NYHA); Edad ≥ 75 años; diabetes mellitus, hipertensión. | Prevención del ictus y de la embolia sistémica en pacientes adultos con fibrilación auricular no valvular, con uno o más factores de riesgo, como por ejemplo, insuficiencia cardiaca congestiva, hipertensión, edad $\geq 75$ años, diabetes mellitus, ictus o ataque isquémico transitorio previos. | Prevención del ictus y de la embolia sistémica en pacientes adultos con fibrilación auricular no valvular, con uno o más factores de riesgo, como por ejemplo, ictus o ataque isquémico transitorio previos, edad ≥ 75 años hipertensión, diabetes mellitus, insuficiencia cardiaca congestiva. |
| Posología habitual | 150 mg BID | 20 mg OD | 5 mg BID |
| Ajuste de dosis | <ul> <li>110 mg BID en:</li> <li>Edad ≥ 80 años.</li> <li>Insuficiencia renal moderada (ACr: 30-49 ml/min) y/o edad 75-79 años cuando el riesgo hemorrágico es alto (ej: peso &lt; 50 kg, AAS, AINE, clopidogrel, etc.)</li> <li>Tratamiento con verapamil.</li> </ul> | 15 mg OD en: - Insuficiencia renal moderada (ACr: 30-49 ml/min). - Insuficiencia renal grave (ACr: 15-29 ml/min). | 2,5 mg BID en: Pacientes con al menos 2 de los 3 siguientes criterios: - Edad ≥ 80 años. - Peso corporal ≤ 60 kg. - Creatinina sérica ≥ 1,5 mg/dl (133 micromol/l) Pacientes con insuficiencia renal grave (ACr: 15-29 ml/min) |
| Contraindicaciones | <ul> <li>Alergia al principio activo o excipientes (colorante amarillo anaranjado E-110).</li> <li>Insuficiencia renal grave (ACr &lt; 30 ml/min).</li> <li>Hemorragia activa clínicamente significativa.</li> <li>Lesión o enfermedad con riesgo significativo de hemorragia mayor.*</li> <li>Tratamiento concomitante con cualquier otro fármaco anticoagulante como la heparina no fraccionada (HNF), heparina de bajo peso molecular (enoxaparina, dalteparina, etc.), fármacos similares a la heparina (fondaparinux, etc.) anticoagulantes orales (ej.: warfarina rivaroxabán, apixabán,), excepto bajo circunstancias de cambio de terapia desde/hacia dabigatrán, o cuando la HNF se da a dosis necesarias para mantener la permeabilidad de un catéter arterial o venoso central.</li> <li>Insuficiencia o enfermedad hepática que pueda afectar a la supervivencia.</li> <li>Administración concomitante con ketoconazol por vía sistémica, ciclosporina, itraconazol, tacrolimus y dronedarona.</li> <li>Pacientes con prótesis valvulares cardiacas</li> </ul> | <ul> <li>Alergia al principio activo o excipientes (lactosa monohidrato).</li> <li>Hemorragia activa clínicamente significativa.</li> <li>Lesión o enfermedad con riesgo significativo de hemorragia mayor.*</li> <li>Tratamiento concomitante con cualquier otro fármaco anticoagulante como la heparina no fraccionada (HNF), heparina de bajo peso molecular (enoxaparina, dalteparina, etc.), fármacos similares a la heparina (fondaparinux, etc.) anticoagulantes orales ((ej.: warfarina, apixabán, dabigatrán), excepto bajo circunstancias de cambio de terapia desde/hacia rivaroxabán, o cuando la HNF se da a dosis necesarias para mantener la permeabilidad de un catéter arterial o venoso central.</li> <li>Hepatopatía asociada a coagulopatía y con riesgo clínicamente relevante de hemorragia, incluidos los pacientes cirróticos con Child Pugh B y C.</li> <li>Embarazo y lactancia.</li> </ul> | <ul> <li>Alergia al principio activo o excipientes (lactosa monohidrato).</li> <li>Hemorragia activa clínicamente significativa.</li> <li>Lesión o enfermedad con riesgo significativo de hemorragia mayor.*</li> <li>Hepatopatía asociada a coagulopatía y con riesgo clínicamente relevante de hemorragia,</li> <li>Tratamiento concomitante con cualquier otro fármaco anticoagulante como la heparina no fraccionada (HNF), heparina de bajo peso molecular (enoxaparina, dalteparina, etc.), fármacos similares a la heparina (fondaparinux, etc.) anticoagulantes orales ((ej.: warfarina, rivaroxabán, dabigatrán), excepto bajo circunstancias de cambio de terapia desde/hacia apixabán, o cuando la HNF se da a dosis necesarias para mantener la permeabilidad de un catéter arterial o venoso central.</li> </ul> |
| Precauciones especiales | Evaluar función renal: - antes de iniciar tratamiento: a fin de excluir pacientes con insuficiencia renal grave (es decir, ACr < 30 ml/min). - durante el tratamiento: como mínimo una vez al año o más frecuentemente si hay sospecha de deterioro renal (ej.: hipovolemia, deshidratación, medicaciones nefrotóxicas). - Estrecha monitorización clínica en situaciones de alto riesgo de sangrado. | <ul> <li>No recomendado en ACr &lt; 15 ml/min ni en<br/>insuficiencia hepática severa.</li> </ul> | <ul> <li>No recomendado en ACr &lt; 15 ml/min ni en insuficiencia hepática severa.</li> <li>Pruebas de función hepática antes de iniciar el tratamiento. Uso con precaución en pacientes con ALT/AST &gt; 2xLSN o bilirrubina total &gt; 1,5xLSN</li> </ul> |

Tabla 1. Condiciones de autorización en la prevención del ictus y embolia sistémica en pacientes con fibrilación auricular no valvular. ACr = aclaramiento de creatinina; BID = dos veces al día (cada 12 horas); OD = una vez al día; \*Lesiones o enfermedades con riesgo significativo de hemorragia mayor: úlcera gastrointestinal actual o reciente, presencia de neoplasias malignas con alto riesgo de sangrado, lesión espinal o cerebral reciente, cirugía espinal u ocular, hemorragia intracraneal reciente, varices esofágicas conocidas o sospechadas, malformaciones arteriovenosas, aneurismas vasculares o anormalidades vasculares intracespinales o intracerebrales importantes.

NOTA: la ficha técnica de los medicamentos puede haber variado desde la publicación de este documento. La ficha técnica actualizada que contiene los últimos cambios incorporados se encuentra disponible en la página web de la AEMPS.

**Dabigatrán (Pradaxa®).** La conclusión sobre el beneficio/riesgo favorable de dabigatrán en la prevención del ictus y la embolia sistémica en pacientes con FA no valvular y al menos un factor de riesgo adicional de complicaciones

tromboembólicas [4,5] deriva principalmente del estudio pivotal RE-LY [22], un ensayo multicéntrico, aleatorizado, abierto, comparativo frente a dosis ajustadas de warfarina para un INR ajustado entre 2-3 (ANEXO I).





Rivaroxabán (Xarelto®). La conclusión sobre el beneficio/riesgo favorable de rivaroxabán en la prevención del ictus y la embolia sistémica en pacientes con FA no valvular y al menos un factor de riesgo adicional de complicaciones tromboembólicas [6,7] deriva principalmente del estudio pivotal ROCKET-AF [23], un ensayo multicéntrico, aleatorizado, dobleciego, comparativo frente a dosis ajustadas de warfarina para un INR ajustado entre 2-3 (ANEXO I).

Apixabán (Eliquis®). La conclusión beneficio/riesgo favorable de apixabán para la prevención del ictus y la embolia sistémica en pacientes con FA no valvular y al menos un factor de riesgo adicional de complicaciones tromboembólicas [8,9] deriva principalmente del estudio pivotal ARISTOTLE) [24], multicéntico, aleatorizado, doble-ciego, comparativo frente a warfarina para un INR ajustado entre 2-3 (ANEXO I). También se evaluaron los datos de un estudio dobleciego, comparativo con ácido acetilsalicílico (AAS) (estudio AVERROES) [25] en la prevención del ictus y embolia sistémica en pacientes con FA cuyos resultados no modificaron la indicación de apixabán pero se encuentran disponibles en el apartado 5.1 de la Ficha Técnica.

No existen estudios que comparen directamente los nuevos anticoagulantes entre sí y existen notables diferencias metodológicas entre los estudios que los comparan con AVK (grado de enmascaramiento, edad y riesgo basal de la población, calidad del control del INR entre otras). Tanto dabigatrán como rivaroxabán y apixabán presentan un perfil beneficio/riesgo favorable para la prevención del ictus y la embolia sistémica en pacientes con FA no valvular y al menos un factor de riesgo adicional de complicaciones tromboembólicas. Todos ellos son alternativas terapéuticas válidas en esta indicación.

#### 2. EVALUACIÓN DEL RIESGO TROMBOEMBÓLICO Y HEMORRÁGICO

La decisión de iniciar o no tratamiento antitrombótico se debe tomar de forma individualizada a partir de la evaluación del riesgo trombótico y hemorrágico en cada paciente.

#### 2.1. Evaluación de riesgo tromboembólico

La escala CHADS<sub>2</sub> [26] es la escala de evaluación de riesgo tromboembólico que dispone de mayor experiencia de uso en la práctica y la más utilizada en la literatura científica (Tabla 2). Existe consenso en las guías internacionales sobre la preferencia de anticoagular, salvo contraindicación, a aquellos pacientes con una puntuación CHADS $_2 \ge 2$  [1,2,27,28], mientras que en pacientes con una puntuación CHADS<sub>2</sub> < 2, la decisión terapéutica debe individualizarse. Más recientemente se ha propuesto la escala CHA<sub>2</sub>DS<sub>2</sub>-VASc [29] que contempla criterios adicionales para discriminar mejor el riesgo embólico de los pacientes con puntuación CHADS<sub>2</sub> < 2. Esta nueva escala ha sido adoptada en las recomendaciones de la Sociedad Europea de Cardiología (ESC) [1], pero no así en recomendaciones análogas de otros países como Estados Unidos [2,27] o Canadá [27]. No existen en la actualidad datos concluyentes de estudios aleatorizados que permitan concluir que la anticoagulación presente una relación beneficio/riesgo superior a la antiagregación con AAS o con AAS y clopidogrel en pacientes con CHADS<sub>2</sub> < 2.

#### 2.2. Evaluación de riesgo hemorrágico

El riesgo de hemorragia se debe valorar en todos los pacientes candidatos a la TAO. La guía europea de FA [1] propone la utilización de la escala HAS-BLED (Tabla 2) [30]. Una puntuación de 3 o más indica un alto riesgo de sangrado.

| CHADS <sub>2</sub> * | Descripción | Puntos |
|---|---|---|
| C ("Congestive heart failure") | historia reciente de insuficiencia cardiaca congestiva | 1 |
| H ("Hypertension") | historia de hipertensión arterial | 1 |
| A ("Age") | edad > 75 años | 1 |
| <b>D</b> ("Diabetes") | historia de diabetes mellitus | I |
| $S_2$ ("Stroke") | historia de ictus/AIT, puntuación doble | 2 |
| Puntuación máxima | | 6 |

| HAS-BLED† | Descripción | Puntos |
|---|---|---|
| H ("Hypertension") | Hipertensión no controlada con presión arterial sistólica ≥ 160 mmHg | 1 |
| A ("Abnormal kidney<br>and/or liver function") | Insuficiencia renal [Diálisis crónica, transplante renal o creatinina sérica ≥ 200 µmol/L (≥ 2,3 mg/dl)] o insuficiencia hepática (cirrosis o datos bioquímicos indicativos de deterioro hepático, BRB > 2 veces el limite superior normal, AST/ALT > 3 veces el límite superior normal, etc.). | 1 ó 2 |
| <b>S</b> ("Stroke") | Historia previa de ictus | 1 |
| B ("Bleeding") | Historia de sangrado, anemia o<br>predisposición al sangrado (ej.: diátesis<br>hemorrágica) | 1 |
| L ("Labile INR") | INR inestable/alto o pobre (menos del<br>60% del tiempo dentro de rango<br>terapéutico) | 1 |
| E ("Elderly") | Edad ≥ 65 años | 1 |
| <b>D</b> ("Drugs and/or alcohol") | Medicamentos que afecten la hemostasia (ej.: $AAS$ , clopidogrel) y/o ingesta de $\geq 8$ bebidas alcohólicas a la semana | 1 ó 2 |
| Puntuación máxima | | 9 |

Tabla 2. Evaluación del riesgo tromboembólico y hemorrágico. \*Gage et al, 2001. †Adaptado de Pisters et al, 2010. AAS = ácido acetilsalicílico; AST/ALT = aspartato-transferasa/alanino-transferasa; AIT = accidente isquémico transitorio; PBP = hiliprophica

La utilización de dicha escala tiene diversas limitaciones. Por una parte, es difícil diferenciar el riesgo embólico del hemorrágico, ya que varios de los factores de riesgo hemorrágico lo son también de riesgo embólico. Por otra parte, de la evaluación del riesgo hemorrágico por la escala HAS-BLED no se derivan recomendaciones terapéuticas más allá de realizar un seguimiento más estrecho en pacientes con alto riesgo hemorrágico.

#### 3. INDICACIÓN DE TRATAMIENTO ANTICOAGULANTE EN PACIENTES CON FIBRILACIÓN AURICULAR NO VALVULAR

Aún aceptando que la decisión de iniciar tratamiento anticoagulante debe individualizarse [1,2,27,28], puede establecerse como regla general que se recomienda la TAO (tradicionalmente con AVK hasta alcanzar un INR estable en un rango de 2-3) en pacientes con una **puntuación CHADS** $_2 \ge 2$ .





#### 4. ELECCIÓN DEL ANTICOAGULANTE EN PACIENTES CON FIBRILACIÓN AURICULAR NO VALVULAR QUE REQUIEREN TRATAMIENTO ANTICOAGULANTE ORAL

Se define la FA no valvular como aquella que no se asocia a estenosis mitral u otra valvulopatía significativa que requiera tratamiento específico programado o ya efectuado (prótesis, valvuloplastia). Considerando los datos de eficacia y seguridad evaluados por las autoridades reguladoras europeas sobre los NACO, las potenciales ventajas e inconvenientes asociados a su uso respecto al de los AVK, la experiencia de uso con cada una de las alternativas terapéuticas, y en los que la anticoagulación se considere indicada (sección 3), se establecen las siguientes recomendaciones para la elección del tipo de anticoagulante:

# 4.1. Situaciones en las que los AVK continúan siendo la opción terapéutica recomendada en el marco del SNS

- Pacientes ya en tratamiento con AVK y buen control de INR. En estos pacientes no se recomienda cambiar a los nuevos anticoagulantes, salvo que exista alguna razón adicional que lo justifique (sección 4.2);
- Nuevos pacientes con fibrilación auricular no valvular en los que esté indicada la anticoagulación. En estos pacientes se recomienda iniciar tratamiento con AVK, salvo que exista algún criterio que justifique iniciar el tratamiento con nuevos anticoagulantes (sección 4.2).
- Fibrilación auricular con afectación valvular, definida como estenosis mitral u otra valvulopatía significativa que requiera tratamiento específico programado o ya efectuado (prótesis, valvuloplastia). Los AVK son de elección. Dabigatrán se encuentra contraindicado en pacientes con prótesis valvulares cardíacas [31].
- 4.2. Situaciones en pacientes con fibrilación auricular no valvular en las que los NACO pueden considerarse una opción terapéutica en el marco del SNS (excluyendo las contraindicaciones generales para la TAO; ver sección 4.3);

#### 4.2.1. Situaciones clínicas:

- Pacientes con hipersensibilidad conocida o con contraindicación específica al uso acenocumarol o warfarina:
- Pacientes con antecedentes de hemorragia intracraneal (HIC) (excepto durante la fase aguda) en los que se valore que los beneficios de la anticoagulación superan el riesgo hemorrágico;
- Pacientes con ictus isquémico que presenten criterios clínicos y de neuroimagen de alto riesgo de HIC, definido como la combinación de HAS-BLED ≥ 3 y al menos uno de los siguientes: leucoaraiosis grado III-IV [32] y/o microsangrados corticales múltiples [33]. Los NACO podrían representar un beneficio en comparación con AVK en estos pacientes debido a su menor potencial para inducir HIC [22,23; ANEXO I];
- Pacientes en tratamiento con AVK que sufren episodios tromboembólicos arteriales graves a pesar de un buen control de INR. Entre otras opciones terapéuticas, los

NACO podrían representar una alternativa en estos pacientes;

#### 4.2.2. Situaciones relacionadas con el control de INR:

- Pacientes que han iniciado tratamiento con AVK en los que no es posible mantener un control de INR dentro de rango (2-3) a pesar de un buen cumplimiento terapéutico. Se considerará que el control de INR es inadecuado cuando el porcentaje de tiempo en rango terapéutico (TRT) sea inferior al 65% [34], calculado por el método de Rosendaal [35]. En los casos en los que este método no esté disponible, se considerará que el control de INR es inadecuado cuando el porcentaje de valores de INR dentro de rango terapéutico sea inferior al 60%. En cualquiera de los supuestos, el periodo de valoración es de al menos los últimos 6 meses, excluyendo los INR del primer mes (en caso de ajuste inicial de dosis) o periodos de cambio debidos a intervenciones quirúrgicas o dentales u otros procedimientos invasivos, etc. que conlleven modificación de la pauta de AVK.
- Imposibilidad de acceso al control de INR convencional.

# 4.3. Situaciones generales en las que la TAO (ya sea con AVK o NACO) está contraindicada o ésta es inconveniente

Algunas de estas circunstancias pueden no corresponder a contraindicaciones absolutas, debiéndose valorar cuidadosamente e individualmente los beneficios y los riesgos de iniciar o suspender la terapia antitrombótica y las posibles alternativas terapéuticas para anticoagulación (p.ej.: utilización de heparinas para anticoagulación durante el embarazo, al menos durante el primer trimestre, ya que los AVK están contraindicados):

- Pacientes que no colaboren y no estén bajo supervisión. Por ejemplo: pacientes con deterioro cognitivo significativo, alcohólicos o con trastornos psiquiátricos, no supervisados.
- Embarazo.
- Hemorragia aguda (al menos durante las 2 primeras semanas tras el episodio), incluyendo hemorragia gastrointestinal, intracraneal, urogenital o del sistema respiratorio, pericarditis aguda, derrames pericárdicos y endocarditis infecciosa.
- Intervenciones quirúrgicas recientes o previstas en el sistema nervioso central.
- Hipertensión grave y/o no controlada.
- Enfermedades hepáticas o renales graves (por el riesgo de sangrado).
- Alteración de la hemostasia (coagulación, fibrinolisis, función plaquetaria) hereditaria o adquirida con riesgo clínicamente relevante de hemorragia: hepatopatía asociada a coagulopatía; diátesis hemorrágica o discrasia sanguínea hemorrágica; trombocitopenias con recuentos plaquetarios inferiores a 50.000/mm3; aumento de la actividad fibrinolítica (p.ej. tras operaciones de pulmón, próstata, útero, etc.); tratamiento concomitante con fibrinolíticos.

Las contraindicaciones de los NACO han sido recientemente actualizadas para incluir una definición homogénea de lesión o enfermedad con riesgo significativo de hemorragia mayor, así





como inclusión de los tratamientos concomitantes con otros antitrombóticos que se consideran contraindicados (Tabla 1).

#### 5. PRECAUCIONES EN EL INICIO Y SEGUIMIENTO DEL TRATAMIENTO ANTICOAGULANTE EN PACIENTES CON FIBRILACIÓN AURICULAR NO VALVULAR

#### 5.1 Inicio del tratamiento

Antes de iniciar el tratamiento se deberán valorar el riesgo tromboembólico y hemorrágico en cada paciente, estableciendo la alternativa terapéutica más adecuada en cada caso. Asimismo, es muy importante evaluar el grado esperable de cumplimiento terapéutico, dado que la falta de cumplimiento podría comprometer la eficacia del tratamiento antitrombótico. Es improbable que un paciente no cumplidor con otras medicaciones lo sea con los NACO.

La decisión de iniciar tratamiento con los NACO debe tomarse tras informar al paciente sobre los riesgos y beneficios del nuevo anticoagulante en comparación con los AVK. Para los pacientes en tratamiento con AVK, se deben considerar los riesgos y beneficios potenciales de cambiar al nuevo anticoagulante teniendo en cuenta su nivel de control de INR.

A la hora de iniciar tratamiento con dabigatrán se deben seguir las recomendaciones recientes de la AEMPS con respecto a la evaluación de la función renal [36]:

- Antes de iniciar el tratamiento debe evaluarse la función renal en todos los enfermos y no debe utilizarse en pacientes con insuficiencia renal grave.
- Durante el tratamiento, debe evaluarse la función renal al menos una vez al año y más frecuentemente en determinadas situaciones clínicas cuando se sospeche que la función renal podría disminuir o deteriorarse.

Como medida general, se recomienda el mismo grado de monitorización de la función renal en el caso de rivaroxabán y apixabán, ya que se requiere ajuste de dosis y/o precaución especial en presencia de insuficiencia renal moderada-grave (Tabla 1). Igualmente, es necesario realizar pruebas de función hepática antes de iniciar el tratamiento con apixabán.

#### 5.2. Seguimiento de los pacientes

En todos los supuestos en los que la TAO esté indicada, se recomienda un seguimiento clínico continuado de los pacientes, evaluando el cumplimiento terapéutico, así como las situaciones clínicas en las que sea necesario interrumpir o ajustar el tratamiento anticoagulante (ej.: aparición de sangrados y/o otros efectos adversos, intervenciones quirúrgicas, ajustes de dosis por variación en la función renal, interacciones farmacológicas u otra causa, cambio del tipo de anticoagulante, etc.) (ANEXO II) [37].

Este seguimiento debe efectuarse con frecuencia. La no necesidad de monitorización rutinaria de la actividad anticoagulante para los NACO no es justificación para relajar el seguimiento clínico. De hecho, dada su menor duración de la acción, las complicaciones tromboembólicas relacionadas con el mal cumplimiento terapéutico podrían ser más frecuentes y tempranas que con los AVK. Se recomienda que dicho seguimiento se efectúe por personal entrenado en el manejo del tratamiento anticoagulante. Se recomienda que los centros

dispongan de protocolos de actuación para el manejo de las complicaciones hemorrágicas, preparaciones para cirugía y exploraciones invasivas en pacientes tratados con los NACO, teniendo en cuenta que no se dispone aún de antídotos específicos para estos nuevos fármacos. Dichos protocolos deben tener en cuenta la información recogida en las fichas técnicas autorizadas de los diferentes medicamentos [4,6,8], así como las guías de práctica clínica disponibles (ANEXO II) [37].

Según las recomendaciones de la ficha técnica las cápsulas de dabigatrán no deben ser almacenadas fuera del envase original, con el objetivo de preservarlas de la humedad, ya que esto puede afectar a la actividad del fármaco. Por lo que, en caso de ser necesario introducirlas en pastilleros, deberá de hacerse con el propio blister recortado.

# 6. CRITERIOS PARA EL USO DE LOS NUEVOS ANTICOAGULANTES

Con el objetivo de orientar la selección de pacientes que serían candidatos a tratamiento, la tabla 3 muestra, en formato de listado, los criterios que debe cumplir un paciente para ser tratado con uno de los NACO, así como su referencia en las secciones anteriores. Para iniciar tratamiento con uno de los NACO, el paciente debe cumplir TODOS los criterios siguientes:

- 1 Presencia de fibrilación auricular NO valvular con indicación de tratamiento anticoagulante (ver sección 3)
- 2 Ausencia de contraindicaciones generales para anticoagulación (ver sección 4.3)
- 3 Presencia de al menos una de las situaciones clínicas que se detallan en las secciones 4.2.1 o 4.2.2.
- 4 Ausencia de contraindicaciones específicas para los nuevos anticoagulantes (ver tabla 1 y referencias 4, 6 y 8)
- 5 Capacidad para entender el riesgo beneficio de la anticoagulación y/o con atención familiar/social que lo entienda
- 6 Historia de buen cumplimiento terapéutico previo que permita prever de forma razonable la buena adaptación a las instrucciones del nuevo tratamiento (ver secciones 5.1 y 5.2)
- 7 Posibilidad fiable de seguimiento periódico de los controles que sean necesarios (clínicos, seguimiento de la función renal; ver sección 5.2)

Tabla 3. Criterios para el uso de los nuevos anticoagulantes. Para que un paciente sea candidato a tratamiento con los nuevos anticoagulantes debe cumplir todos los criterios anteriores.

#### 7. NOTIFICACIÓN DE REACCIONES ADVERSAS

Se recuerda a los profesionales sanitarios la necesidad de notificar las sospechas de reacciones adversas, en particular por tratarse de fármacos de reciente comercialización. Todas las sospechas de reacciones adversas atribuidas al medicamento serán notificadas a través de la tarjeta amarilla a los Centros de Farmacovigilancia de cada Comunidad Autónoma.

Para mayor información sobre notificación de reacciones adversas, se puede consultar la web de la AEMPS: <a href="http://www.aemps.gob.es/vigilancia/medicamentosUsoHumano/docs/notificacion-SRA.pdf">http://www.aemps.gob.es/vigilancia/medicamentosUsoHumano/docs/notificacion-SRA.pdf</a>

#### 8. REFERENCIAS

1. Camm AJ, Kirchhof P, Lip GY, et al. Guidelines for the management of atrial fibrillation: the Task Force for the Management of





Atrial Fibrillation of the European Society of Cardiology (ESC). Eur Heart J. 2010; 31: 2369-429.

- 2. Furie KL, Kasner SE, Adams RJ, et al. Guidelines for the Prevention of Stroke in Patients With Stroke or Transient Ischemic Attack: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2011; 42: 227-76
- 3. Cea-Calvo L, Redón J, Lozano JV, et al. Prevalencia de fibrilación auricular en la población española de 60 o más años de edad. Estudio PREV-ICTUS. Rev Esp Cardiol. 2007; 60: 616-24.
- 4. Pradaxa® Ficha Técnica. Disponible en: <a href="www.aemps.gob.es">www.aemps.gob.es</a> (CIMA).
- 5. CHMP assessment report. Pradaxa® procedure No. EMEA/H/C/000829/X/13/G. Doc. Ref.: EMA/CHMP/203468/2011. London, 23 August 2011. Disponible en: <a href="http://www.ema.europa.eu/docs/en\_GB/document\_library/EPAR\_-">http://www.ema.europa.eu/docs/en\_GB/document\_library/EPAR\_-</a> Assessment Report Variation/human/000829/WC500110875.pdf
- 6. Xarelto® Ficha Técnica. Disponible en: <a href="www.aemps.gob.es">www.aemps.gob.es</a> (CIMA)
- 7. CHMP assessment report. Xarelto® procedure EMEA/H/C/000944/II/0012. Doc. Ref: EMA/42547/2012. London, 20 January 2012. Disponible en: <a href="http://www.ema.europa.eu/docs/en\_GB/document\_library/EPAR">http://www.ema.europa.eu/docs/en\_GB/document\_library/EPAR</a> -

Assessment Report - Variation/human/000944/WC500120735.pdf

- 8. Eliquis® Ficha Técnica. Disponible en: <a href="www.aemps.gob.es">www.aemps.gob.es</a> (CIMA)
- 9. CHMP assessment report. Eliquis® procedure No. EMEA/H/C/002148/X/0004/G. Doc. Ref.: EMA/XXX. London, X November 2012. Disponible en: XXX (Pending EC decision)
- 10. Gómez D, Paladio N, Almazán C; Agència d'Informació, Avaluació i Qualitat en Salut. Servei Català de la Salut. Departament de Salut. Generalitat de Catalunya, Dabigatrán etexilat en la profilaxi de l'accident vascular cerebral i de l'embolisme sistèmic en fibril·lació auricular no valvular. Noviembre 2011. Disponible en: <a href="http://www10.gencat.cat/catsalut/archivos/instruccions/instruccio\_03-2011">http://www10.gencat.cat/catsalut/archivos/instruccions/instruccio\_03-2011</a> informe dabigatrán.pdf
- 11. Baquero Barroso MJ, Álvarez-Cienfuegos A, Candela Marroquín E; Oficina de Evaluación de Medicamentos. Servicio Extremeño de Salud. Dabigatrán [en fibrilación auricular no valvular]. Hoja de Evaluación de Nuevos Medicamentos. 2011;(2). Disponible en: <a href="http://saludcomunitaria.files.wordpress.com/2011/11/20110930-deofevalmto-hnft-dabigatrc3a1n-fa-v10.pdf">http://saludcomunitaria.files.wordpress.com/2011/11/20110930-deofevalmto-hnft-dabigatrc3a1n-fa-v10.pdf</a>
- 12. Grupo de Trabajo; Subdirección General de Compras de Farmacia y Productos Sanitarios de la Consejería de Sanidad de la Comunidad de Madrid. Nuevos anticoagulantes para la prevención del ictus en la fibrilación auricular no valvular: Recomendaciones de la Comunidad de Madrid. Diciembre 2011. Disponible en: <a href="http://www.madrid.org/cs/">http://www.madrid.org/cs/</a>
- 13. SACYL. Dabigatrán: pros y contras. Disponible en: <a href="http://www.fqscyl.es/profesionales/es/farmacia/uso-racional-medicamento/publicaciones-urm/dabigatran-pros-contras">http://www.fqscyl.es/profesionales/es/farmacia/uso-racional-medicamento/publicaciones-urm/dabigatran-pros-contras</a>
- 14. Servicio de Uso Racional del Medicamento. Dirección General de Farmacia. Servicio Canario de Salud. Indicación revisada del Dabigatrán (Pradaxa®). Diciembre 2011. Disponible en: <a href="http://www2.gobiernodecanarias.org/sanidad/scs/content/b6c8828b-2701-1e1-bded-83400f7d5093/Noticia\_Indicaci%C3%B3n\_%20revisada\_Dabigatran.pdf">http://www2.gobiernodecanarias.org/sanidad/scs/content/b6c8828b-2701-1e1-bded-83400f7d5093/Noticia\_Indicaci%C3%B3n\_%20revisada\_Dabigatran.pdf</a>
- 15. Galindo Rueda MM. Dabigatrán. Fibrilación auricular no valvular. Hoja de evaluación de medicamentos. Octubre 2011, Vol. XII(2). Disponible en:
- $\underline{http://www.murciasalud.es/recursos/ficheros/223029\text{-}dabigatran.pdf}$
- 16. Resolución 291/2012, de 10 de febrero, del Director Gerente del Servicio Navarro de Salud-Osasunbidea, por la que se aprueban

- instrucciones para la utilización de Dabigatrán (PRADAXA®) en el Servicio Navarro de Salud-Osasunbidea.
- 17. Osakidetza. Dabigatrán (Pradaxa) en el tratamiento de la fibrilación auricular no valvular. INFAC. Vol. 20(1). 2012. Disponible en: <a href="http://www.osakidetza.euskadi.net/r85-ckpubl02/eu/contenidos/informacion/cevime\_infac/eu\_miez/adjuntos/Infac\_Vol\_20\_n\_1.pdf">http://www.osakidetza.euskadi.net/r85-ckpubl02/eu/contenidos/informacion/cevime\_infac/eu\_miez/adjuntos/Infac\_Vol\_20\_n\_1.pdf</a>
- 18. Agencia de Evaluación de Tecnologías Sanitarias de Andalucía (AETSA). Nuevos anticoagulantes orales para la prevención del ictus y la embolia sistémica en fibrilación auricular no valvular. Septiembre 2012.Disponible en:
- http://www.juntadeandalucia.es/salud/servicios/contenidos/nuevaaetsa/up/AETSA\_2012-2\_ACOs\_def.pdf
- 19. Agencia de Evaluación de Tecnologías Sanitarias de Andalucía (AETSA).Guía para la elección de tratamiento anticoagulante oral en la prevención de las complicaciones tromboembólicas asociadas a la fibrilación auricular no valvular. Octubre 2012. Disponible en: http://www.guiasalud.es/GPC/GPC\_517\_Tratamiento%20anticoagulante\_guia\_rapida.pdf
- 20. Hart RG, Pearce LA, Aguilar MI. Meta-analysis: Antithrombotic therapy to prevent stroke in patients who have nonvalvular atrial fibrillation. Ann Intern Med. 2007: 146: 857-67.
- 21. Navarro JL, César JM, Fernández MA, et al. Tratamiento anticoagulante oral. Estudio coste/beneficio. Rev Adm Sanit. 2008; 6: 525-42.
- 22. Connolly SJ, Ezekowitz MD, Yusuf S, et al. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009; 361: 1139-51
- 23. Patel MR, Mahaffey KW, Garg J, et al. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011; 365: 883-
- 24. Granger CB, Alexander JH, McMurray JJ, et al. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011; 365: 981-92
- 25. Connolly SJ, Eikelboom J, Joyner C, et al. Apixaban in patients with atrial fibrillation. N Engl J Med. 2011; 364: 806-17.
- 26. Gage BF, Waterman AD, Shannon W, et al. Validation of clinical classification schemes for predicting stroke: results from the national registry of atrial fibrillation. JAMA. 2001; 285: 2864-70.
- 27. You JJ, Singer DE, Howard PA, et al. Antithrombotic therapy for atrial fibrillation: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012; 141(2 Suppl): e531S-75S.
- 28. Skanes AC, Healey JS, Cairns JA, et al; Canadian Cardiovascular Society Atrial Fibrillation Guidelines Committee. Focused 2012 update of the Canadian Cardiovascular Society atrial fibrillation guidelines: recommendations for stroke prevention and rate/rhythm control. Can J Cardiol. 2012; 28: 125-36.
- 29. Lip GY, Nieuwlaat R, Pisters R, et al. Refining clinical risk stratification for predicting stroke and thromboembolism in atrial fibrillation using a novel risk factor-based approach: The Euro Heart Survey on Atrial Fibrillation. Chest. 2010; 137: 263–72.
- 30. Pisters R, Lane DA, Nieuwlaat R, et al. A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest. 2010; 138: 1093-100
- 31. Agencia Española de Medicamentos y Productos Sanitarios. Dabigatrán (Pradaxa®): contraindicación en pacientes con prótesis valvulares cardíacas. Diciembre 2012. Disponible en:http://www.aemps.gob.es/informa/notasInformativas/medicamentosUs oHumano/seguridad/2012/NI-MUH\_FV\_17-2012-dabigatran.htm





- 32. Smith EE, Rosand J, Knudsen KA, et al. Leukoaraiosis is associated with warfarin-related hemorrhage following ischemic stroke. Neurology. 2002; 59: 193-7.
- 33. Lee SH, Ryu WS, Roh JK. Cerebral microbleeds are a risk factor for warfarin-related intracerebral hemorrhage. Neurology. 2009; 72: 171-6.
- 34. Connolly SJ, Pogue J, Eikelboom J, et al; ACTIVE W Investigators. Benefit of oral anticoagulant over antiplatelet therapy in atrial fibrillation depends on the quality of international normalized ratio control achieved by centers and countries as measured by time in therapeutic range. Circulation. 2008; 118: 2029-37.
- 35. Rosendaal FR, Cannegieter SC, van der Meer FJ, et al. A method to determine the optimal intensity of oral anticoagulant therapy. Thromb Haemost. 1993; 69: 236-9.
- 36. Agencia Española de Medicamentos y Productos Sanitarios. Dabigatrán (Pradaxa®) y riesgo de hemorragia: nuevas recomendaciones de vigilancia de la función renal. Octubre 2011. Disponible en: <a href="http://www.aemps.gob.es/informa/notasInformativas/medicamentosUsoHumano/seguridad/2011/docs/NI-MUH\_21-2011.pdf">http://www.aemps.gob.es/informa/notasInformativas/medicamentosUsoHumano/seguridad/2011/docs/NI-MUH\_21-2011.pdf</a>
- 37. Guía SEHH-SETH para el manejo de los nuevos anticoagulantes orales. Diciembre 2012. Disponible en: <a href="http://www.sehh.es/documentos\_detalle.php?id=53">http://www.sehh.es/documentos\_detalle.php?id=53</a>

#### **GRUPO DE EXPERTOS**

(por orden alfabético)

#### Laila Abdel-Kader Martín

Agencia de Evaluación de Tecnologías Sanitarias de Andalucía (AETSA). Consejería de Salud. Junta de Andalucía. Sevilla.

#### Cristina Avendaño Solá

Servicio de Farmacología Clínica. Hospital Puerta de Hierro. Madrid.

#### Gonzalo Calvo Rojas

Servicio de Farmacología Clínica. Hospital Clínic. Barcelona.

#### Antoni Dávalos Errando

Departamento de Neurociencias. Hospital Germans Trias i Pujol. Badalona.

#### Cristina Espinosa Tomé

Gerència d'Atenció Farmacèutica i Prestacions Complementàries. Servei Català de la Salut. Barcelona.

#### **Antonio Gómez-Outes**

División de Farmacología y Evaluación Clínica. Agencia Española de Medicamentos y Productos Sanitarios. Madrid

#### José María Lobos Bejarano

Centro de Salud Jazmín. Madrid.

#### José Luis López-Sendón

Servicio de Cardiología. Hospital de La Paz. Madrid.

#### Pascual Marco Vera

Servicio de Hematología Y Hemoterapia. Hospital General Universitario. Alicante

#### Teresa Molina López

Agencia de Evaluación de Tecnologías Sanitarias de Andalucía (AETSA). Consejería de Salud. Junta de Andalucía. Sevilla.

#### Núria Paladio Duran

Agència d'Informació, Avaluació i Qualitat en Salut (AIAQS). Barcelona

#### Concepción Prieto Yerro

Comité de Medicamentos de Uso Humano (CHMP) de la EMA. Agencia Española de Medicamentos y Productos Sanitarios. Madrid.

#### José Santaló Rios

Centro de Información de Medicamentos. Subdirección Xeral de Farmacia. Servizo Galego de Saúde. Santiago de Compostela

Todos los expertos han realizado una declaración de conflictos de interés.







| Estudio y Referencia | Diseño y objetivo, validez interna | Población estudiada | Pauta de tratamiento | Variables principales de eficacia y seguridad | Resultados |
|---|---|---|---|---|---|
| RE-LY Pradaxa EPAR EMEA/H/C/000829/ X/13/G Connolly, et al. NEJM. 2009; 361: 1139-51. | Diseño: ECA, prospectivo, multicéntrico, de no-inferioridad, doble ciego para grupos DE, abierto grupo WA. Objetivo: comparar la eficacia y seguridad de DE (dos dosis, ambas a doble ciego) respecto a WA (abierto, no ciego) en pacientes con FA y riesgo aumentado de ACV. Validez interna: Estudio abierto, no ciego, lo que limita su validez interna. Análisis de no-inferioridad en la población ITT en lugar de en la población PP, aunque análisis "post-hoc" PP fue consistente con en análisis ITT. | Sujetos aleatorizados: N = 18.113 pacientes Media de edad: 71 años. Varones: 64% DE 150 mg (n=6.076) - DE 110 mg (n=6.015) - WA dosis ajustada (INR: 2-3) (n=6022) Criterios de inclusión: FA y al menos uno de los siguientes: ACV o AIT previo; FEVI <40%; ICC clase funcional ≥ II de la NYHA; edad ≥ 75 años o 65-74 en caso de DM, HTA o enfermedad coronaria. Criterios principales de exclusión (14 en total): Ictus reciente (14 días) o ictus severo (6 meses antes); riesgo aumentado de hemorragia; ACr <30 ml/mir, enfermedad hepática, enfermedad valvular significativa, embarazo. | Tratamientos: - DE 150 mg BID - DE 110 mg BID - WA (dosis ajustada; INR: 2-3) Duración: 2 años (mediana de seguimiento) | Eficacia: Incidencia combinada de ACV y ES. Criterio de no inferioridad: limite superior del IC 95% bilateral (97,5% unilateral) del riesgo relativo de ACV o ES con DE comparado con WA < 1,46. Todos los análisis (no-inferioridad y superioridad) por ITT. Tiempo hasta el primer evento. Modelo de regresión de Cox. Seguridad: Hemorragia mayor (descenso Hb ≥ 20 g/L, transfusión 2 unidades sanguíneas, o hemorragia fatal o en órgano crítico). | ACV/ES: DE 150 mg BID vs. WA (ITT): % anual: 1,11% vs. 1,71% HR: 0,65; IC95%: 0.52 a 0,81 P no-inferioridad ≤ 0,0001 P superioridad = 0,0001 DE 110 mg BID vs. WA (ITT): % anual: 1,54% vs. 1,71% HR: 0,90; IC95%: 0,74 a 1,10 P no-inferioridad ≤ 0,0001 P superioridad = 0,2943 Mortalidad por cualquier causa: DE 150 mg BID vs. WA: % anual: 3,64% vs. 4,13% HR: 0,88; IC95%: 0,77 a 1,00 P superioridad = 0,0517 DE 110 mg BID vs. WA: % anual: 3,75% vs. 4,13% HR: 0,91; IC95%: 0,80 a 1,03 P superioridad = 0,1308 Hemorragia mayor: DE 150 mg BID vs. WA: % anual: 3,32% vs. 3,57% HR: 0,91; IC95%: 0,81 a 1,07 P superioridad = 0,3146 DE 110 mg BID vs. WA: % anual: 3,25%: 0,357% HR: 0,80; IC95%: 0,70 a 0,93 P superioridad = 0,3146 DE 110 mg BID vs. WA: % anual: 3,75% vs. 3,57% HR: 0,80; IC95%: 0,70 a 0,93 P superioridad = 0,0026 Otros: reducción significativa de HIC (RAR ≈ -0,5% anual) y con hemorragia con amenaza para la vida (RAR ≈ -0,5% anual) con ambas dosis de DE, pero aumento significativo de hemorragia GI (RAR ≈ +0,5% anual; dosis de 150 mg BID) y dispepsia (RAR ≈ +3% anual), y tendencia no significativa a más IM (RAR ≈ +0,2% anual) |
| ROCKET-AF<br>Xarelto EPAR<br>EMEA/H/C/000944/<br>II/0012<br>Patel, et al. NEJM. 2011; 365:<br>883-91. | Diseño: ECA, prospectivo, multicéntrico, de no-inferioridad, doble ciego. Objetivo: comparar la eficacia y seguridad de RIV respecto a WA en pacientes con FA y riesgo aumentado de ACV. Validez interna: Estudio doble-ciego. Análisis de no-inferioridad en la población PP. Análisis de superioridad por ITT con disminución del efecto con respecto al análisis PP. | Sujetos aleatorizados: N = 14.264 pacientes Mediana de edad: 73 años. Varones: 60%. - RIV 20 mg (n=7.131) - WA dosis ajustada (INR: 2-3) (n=7.133) Criterios de inclusión: FA con riesgo moderado/alto de ictus (puntuación CHADS₂ ≥ 2): historia de ACV, AIT o ES previo, o al menos 2 de los siguientes factores de riesgo: ICC o FEVI ≤35%; HTA; edad ≥ 75 años; DM. Criterios principales de exclusión (31 en total): Ictus reciente (14 días) o ictus severo (6 meses antes); riesgo aumentado de hemorragia; ACr <30 ml/min; enfermedad hepática, enfermedad valvular significativa, embarazo. | Tratamientos: - RIV 20 mg OD. Reducción de dosis a 15 mg OD si ACr 15-49 ml/min (IR moderada-grave) WA (dosis ajustada; INR:2-3) Duración: 590 días (mediana de seguimiento PP) (707 días ITT) | Eficacia: Incidencia combinada de ACV y ES. Criterio de no inferioridad: límite superior del IC 95% bilateral (97,5% unilateral) del riesgo relativo de ACV o ES con RIV comparado con WA < 1,46. Análisis de no-inferioridad PP y superioridad ITT. Tiempo hasta el primer evento. Modelo de regresión de Cox. Seguridad: Hemorragia clínicamente relevante: incidencia combinada de hemorragia mayor (descenso Hb ≥ 20 g/L, transfusión 2 unidades sanguíneas, o hemorragia fatal o en forgano crítico o incapacidad permanente) y menor clínicamente relevante (no cumple criterios de hemorragia mayor pero requiere atención médica). | ACV/ES: RIV 20 mg OD vs. WA (No-inferioridad PP) % anual: 1,71% vs. 2,16% HR: 0,79; IC95%: 0,66 a 0,96 P no-inferioridad < 0,001 RIV 20 mg OD vs. WA (Superioridad ITT) % anual: 2,12% vs. 2,42% HR: 0,88; IC95%: 0,74 a 1,03 P superioridad = 0,117 Mortalidad por cualquier causa: RIV 20 mg OD vs. WA: % anual: 4,52% vs. 4,91% HR: 0,92; IC95%: 0,82 a 1,03 P superioridad = 0,152 Hemorragia clinicamente relevante: RIV 20 mg OD vs. WA: % anual: 14,91% vs. 14,52% HR: 1,03; IC95%: 0,96 a 1,11 P superioridad = 0,442 Hemorragia mayor: RIV 20 mg OD vs. WA: % anual: 3,60% vs. 3,45% HR: 1,04; IC95%: 0,90 a 1,20 P superioridad = 0,576 Otros: reducción significativa de HIC (RAR ≈ -0,3% anual) y hemorragia fatal (RAR ≈ -0,2% anual) con RIV, pero aumento significativo de hemorragia GI (RAR ≈ -0,2% anual) con RIV, pero aumento significativo de hemorragia GI |



| ARISTOTLE Eliquis® EPAR EMEA/H/C/002148/X/0004/G . Granger et al. NEJM 2011; 365: 981-92. | Diseño: ECA, prospectivo, multicéntrico, de no-inferioridad, doble ciego. Objetivo: comparar la eficacia y seguridad de API respecto a WA en pacientes con FA y riesgo aumentado de ACV. Validez interna: Estudio doble-ciego. | Sujetos aleatorizados: N = 18.201 pacientes Mediana de edad: 70 años. Varones: 65%. - API 5 mg BID (n=9.120) - WA dosis ajustada (INR: 2-3) (n=9.081) Criterios de inclusión: | Tratamientos: - 5 mg BID. Reducción de dosis a 2,5 mg BID en pacientes con al menos 2 de los 3 criterios siguientes: 1) Edad ≥ 80 años; 2) Peso corporal ≤ 60 kg; 3) Creatinina sérica ≥ 1,5 mg/dl (133 | Eficacia: Incidencia combinada de ACV y ES. Criterio de no inferioridad: límite superior del IC 95% bilateral (97,5% unilateral) del riesgo relativo de ACV o ES con RIV comparado con WA < 1,38. Análisis de no-inferioridad y | ACV/ES: API 5 mg BID vs. WA (No-inferioridad y superioridad ITT) % anual: 1,27% vs. 1,60% HR: 0,79; IC95%: 0,66 a 0,95 P no-inferioridad < 0,001 P superioridad = 0,01 Mortalidad por cualquier causa: |
|---|---|---|---|---|---|
| | Análisis de no-inferioridad y superioridad en la población ITT. Análisis secundario PP consistente con el análisis ITT. | FA permanente o persistente con riesgo moderado/alto de ictus (puntuación CHADS₂≥2): edad≥75 años; historia de ACV, AIT o ES previo; ICC sintomática en los últimos 3 meses o FEVI ≤40%; DM; HTA en tto farmacológico. Criterios principales de exclusión (19 en total): AF debida a causas reversibles; estenosis mitral clinicamente significativa o prótesis mecánica; riesgo aumentado de hemorragia; hemorragia intracraneal previa; ACr <25 ml/min; ALT o AST >2×LSN o bilirrubina total≥1,5×LSN | micromol/l) - WA (dosis ajustada; INR:2-3) <b>Duración:</b> 1,8 años (mediana de seguimiento ITT) | superioridad ITT. Tiempo hasta el primer evento. Modelo de regresión de Cox. Seguridad: - Hemorragia mayor (descenso Hb ≥ 20 g/L, transfusión 2 unidades sanguíneas, o hemorragia fatal o en órgano crítico). | API 5 mg BID vs. WA: % anual: 3,52% vs. 3,94% HR: 0,89; IC95%: 0,80 a 0,99 P superioridad = 0,047 Hemorragia mayor: API 5 mg BID vs. WA: % anual: 2,13% vs. 3,09% HR: 0,69; IC95%: 0,60 a 0,80 P superioridad < 0,001 Otros: reducción significativa de HIC (RAR ≈ -0,5% anual) y hemorragia clínicamente relevante (RAR ≈ -1,94% anual) con API, sin diferencias significativas en hemorragia GI. |

ACr = aclaramiento de creatinina; ACV = accidente cerebrovascular; AIT = accidente isquémico transitorio; ALT = alanino-transferasa; API = apixabán; AST = aspartato-transferasa; BID = dos veces al día; DE = dabigatrán etexilato; DM = diabetes mellitus; ECA = ensayo clínico aleatorizado; ES = embolismo sistémico; FA = fibrilación auricular; FEVI = fracción de eyección del ventrículo izquierdo; GI = gastrointestinal; HIC = hemorragia intracraneal; HR = "hazard ratio"; HTA = hipertensión arterial; IC = intervalo de confianza; ICC = insuficiencia cardiaca congestiva; IM = infarto de miocardio; INR = cociente internacional normalizado; ITT = intención de tratar; LSN = limite superior de la normalidad; NYHA = "New York Heart Association"; OD = una vez al día; PP = por protocolo; RAR = reducción absoluta del riesgo; RIV = rivaroxabán; tto = tratamiento; WA = warfarina.





# ANEXO II: Consideraciones prácticas sobre el manejo de las complicaciones hemorrágicas y actitud perioperatoria con los nuevos anticoagulantes orales (NACO) [Basado en referencias 4, 6, 8 y 35].

#### MANEJO DE LAS COMPLICACIONES HEMORRÁGICAS DE LOS NACO

La experiencia del manejo de las complicaciones hemorrágicas de los NACO es escasa. Las recomendaciones generales no difieren de los protocolos de actuación ante una hemorragia secundaria a un fármaco antitrombótico, ya que no disponemos de ningún antídoto específico que neutralice la acción de los NACO.

| Pradaxa (dabigatrán) | Xarelto (rivaroxabán) | Eliquis (apixabán) |
|---|---|---|
| No antidoto específico disponible | No antidoto específico disponible | No antídoto específico disponible |
| Discontinuación del tto | Discontinuación del tto | Discontinuación del tto |
| Investigación/tratamiento del<br>origen del sangrado y medidas<br>generales (e.j.: mediante<br>hemostasia quirúrgica y<br>reemplazo del volumen<br>sanguíneo). | Investigación/tratamiento del origen del sangrado y medidas generales (e.j.: mediante compresión mecánica, intervenciones quirúrgicas, reemplazo hidrico y apoyo hemodinámico, y transfusión de hemoderivados o componentes hemáticos). | Investigación/tratamiento<br>del origen del sangrado y<br>medidas generales (ej.:<br>hemostasia quirúrgica y/o<br>transfusión de plasma<br>fresco). |
| Dado que el dabigatrán se<br>elimina principalmente por vía<br>renal, debe mantenerse una<br>diuresis adecuada. | Puede considerarse el uso<br>de carbón activado para<br>reducir la absorción en caso<br>de sobredosis por<br>rivaroxabán. | La administración de carbón activado tras la ingestión de apixabán entre 2 y 6 h redujo la exposición al fármaco entre un 50% y 27%, respectivamente, y la vida media disminuyó a 5,3 h y 4,9 h, respectivamente. |
| Si el sangrado amenaza la vida del paciente y no puede controlarse con las medidas anteriores, se puede considerar el uso de concentrados del complejo de protrombina activado (p. ej. FEIBA), Factor VIIa recombinante o concentrados de los factores de la coagulación II, IX y X. Hay cierta evidencia experimental que apoya el papel de estos agentes en revertir el efecto anticoagulante de dabigatrán, pero los datos sobre su utilidad en términos clínicos y también sobre el posible riesgo de un tromboembolismo de rebote son muy limitados. | Si el sangrado amenaza la vida del paciente y no puede controlarse con las medidas anteriores, se puede considerar la administración de factor VIIa recombinante. No obstante, no hay experiencia clínica con el uso de factor VIIa y rivaroxabán | Si el sangrado amenaza la vida del paciente y no puede controlarse con las medidas anteriores, se puede considerar la administración de factor VIIa recombinante. No obstante, no hay experiencia clínica con el uso de factor VIIa y apixabán. |
| Se debe considerar la<br>administración de concentrados<br>de plaquetas en caso de<br>trombocitopenia o cuando se<br>hayan utilizado medicamentos<br>antiagregantes de acción<br>prolongada.y otros | No se espera que el sulfato de protamina y la vitamina K afecten a la actividad anticoagulante de rivaroxabán. No hay una justificación cientifica sobre la ventaja ni la experiencia con hemostáticos sistémicos (por ejemplo, desmopresina, aprotinina, ácido tranexámico, ácido aminocaproico) en las personas que reciben rivaroxabán. | |

Dado que la unión a proteínas es baja, el dabigatrán es dializable. Debido a su elevada fijación a las proteínas plasmáticas, no se espera que el rivaroxabán sea dializable.

Tabla II.1. Fuente: Fichas técnicas autorizadas (sección 4.9) de Pradaxa, Xarelto y Eliquis.

En la tabla de la izquierda (tabla II.1) se detallan las recomendaciones establecidas en las fichas técnicas autorizadas de los NACO en caso de sobredosis y/o sangrado.

#### RECOMENDACIONES PARA EL MANEJO DE LAS COMPLICACIONES HEMORRÁGICAS DE LOS NACO

- 1. Evaluación de la gravedad y localización de la hemorragia.
  - 2. Discontinuación del anticoagulante.
- **3. Tratamiento de soporte**: carbón activado (disminución de la absorción del NACO en las primeras 6 horas tras su administración oral); control hemodinámico (repleción de volumen, transfusión, ionotrópicos); localización de la hemorragia y corrección quirúrgica/endoscópica si procede.
- **4. Hemodiálisis** / **hemoperfusión:** sólo válida para dabigatrán, debido a su baja unión a proteínas plasmáticas.
- **5. Administración de procoagulantes:** sólo en casos de amenaza para la vida, ya que pueden asociarse a trombosis.
  - Dabigatrán: concentrados del complejo de protrombina activado (p. ej. FEIBA), Factor VIIa recombinante o concentrados de los factores de la coagulación II, IX y X.
  - Rivaroxabán y apixabán: Factor VIIa recombinante.

#### MANEJO PERIOPERATORIO DE LOS NACO

#### Reversión antes de la cirugía

El efecto de los NACOs es de más corta duración que el de los dicumarínicos y aparece a partir de las 2 horas de su administración oral, siempre que la absorción intestinal no esté alterada. Los datos disponibles señalan que se puede establecer un período de tiempo de seguridad previo a la intervención, sin necesidad de control biológico, teniendo en cuenta la función renal del paciente y el tipo de cirugía (Tabla II-2).

Solo en caso de hemorragia significativa con amenaza vital se considerará el complejo de protrombina activado o el factor VIIa, ya que su uso no está exento de riesgo trombótico.

#### Elección del tipo de anestesia

En situaciones quirúrgicas de urgencia sólo podría contemplarse la opción de anestesia epidural o espinal cuando exista un alto grado de certeza de ausencia de actividad anticoagulante. En los casos de cirugía programada, para la práctica de anestesia locorregional se deberán respetar los siguientes intervalos de tiempo (Tabla II-3).





| ClCr | Vida media (h.) | Tiempo dosis previa.<br>Riesgo bajo de<br>sangrado <sup>b</sup> | Tiempo dosis previa.<br>Riesgo moderado-alto de<br>sangrado |
|---|---|---|---|
| Pradaxa (dabigat | rán) <sup>a</sup> | | |
| >80 ml/min. | 13 | 24 horas | 2 días |
| >50 ≤80<br>ml/min. | 15 | 24 horas | 3 días |
| >30 ≤50<br>ml/min. | 18 | Al menos 2 días | 4 días |
| ≤30 ml/min.<br>(contraindicado) | 27 | 2-4 días | >5 días |
| Xarelto (rivaroxa | bán) | | |
| >30 ml/min. | 7 a 11 | 24 horas | 2 días |
| <30 ml/min. | Desconocido | 2 días | 4 días |
| Eliquis (apixabán) | | | |
| >30 ml/min | 12 | ≥ 24 horas | ≥ 48 horas |
| <30 ml/min | Desconocido | Desconocido | Desconocido |

Tabla II-2. Reversión en cirugía según función renal y riesgo hemorrágico quirúrgico. CICr = aclaramiento de creatinina. a. Para interrupciones del tratamiento inferiores a las 48 horas no es preciso instaurar terapia puente con heparina. b. En situaciones de muy bajo riesgo puede ser suficiente suspender la dosis de la noche anterior y reanudar el tratamiento inmediatamente después del procedimiento. Fuente: Documento de la SETH/SEHH sobre nuevos anticoagulantes orales y fichas técnicas autorizadas de Pradaxa, Xarelto y Eliquis.

# Reintroducción de la anticoagulación a largo plazo tras cirugía

En un paciente en tratamiento a largo plazo con NACO (por ejemplo: fibrilación auricular no valvular) que ha sido intervenido quirúrgicamente, la reanudación del tratamiento con el nuevo anticoagulante tras la cirugía deberá instaurarse tan pronto como sea posible, supuesto que se haya establecido una adecuada hemostasia. En procedimientos con buena hemostasia, se puede reanudar el tratamiento a las 4-6 horas de la cirugía. En el caso de cirugía abdominal mayor o urológica se debe esperar a que no haya hemorragia activa por los drenajes.

| | Pradaxa<br>(dabigatrán) | Xarelto<br>(rivaroxabán) | Eliquis<br>(apixabán) |
|---|---|---|---|
| Tiempo entre inserción o<br>retirada del catéter y<br>(siguiente) dosis del<br>anticoagulante <sup>a</sup> | ≥ 2 horas | ≥ 6 horas (24 horas<br>en caso de punción<br>traumática) | ≥ 5 horas |
| Tiempo entre última<br>dosis del anticogulante e<br>inserción o retirada del<br>catéter | No especificado<br>en la ficha técnica.<br>Al menos 2 vidas<br>medias* (≥ 26<br>horas) | ≥ 18 horas | 20-30 horas |

Tabla II-3. Intervalos de tiempo a tener en cuenta cuando se utiliza la anestesia espinal y tromboprofilaxis con los nuevos anticoagulantes en artroplastia de cadera o rodilla. Fuente: richas Técnicas autorizadas de Pradaxa, Xarelto y Eliquis; \*Rosencher et al. 2007. a. Si existe una punción traumática, la siguiente/primera dosis del anticoagulante se debe retrasar 24 horas.

#### RECOMENDACIONES PARA EL MANEJO PERIOPERATORIO DE LOS NACO

- 1. En todo paciente se debe evaluar el riesgo hemorrágico de la intervención, así como la función renal.
- 2. Es fundamental conocer cuándo se administró la última dosis.

- 3. En cirugía programada, se recomienda esperar al menos 24 h en caso de riesgo hemorrágico bajo y al menos 48 h en caso de riesgo hemorrágico moderado-alto.
- 4. En cirugía urgente, se recomienda esperar al menos 12 h tras la última dosis si es posible, y se deberá optar habitualmente por anestesia general.
- 5. Solo en caso de hemorragia significativa con amenaza vital se considerará el concentrado de complejo protrombínico o factor VIIa, ya que su uso no está exento de riesgo trombótico.
- 6. En caso de anestesia espinal concomitante, se deberán respetar unos tiempos mínimos entre inserción/retirada del catéter y dosis del anticoagulante.
- 7. La reanudación del tratamiento con el nuevo anticoagulante tras la cirugía deberá instaurarse tan pronto como sea posible, siempre que se haya establecido una adecuada hemostasia.



#### APPROVAL / SIGNATURE PAGE

Document Number: c09057375 Technical Version Number: 1.0

Document Name: non-interventional-study-protocol-spain-version-01

Title: non-interventional-study-protocol-spain-version-01

#### **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | Date Signed |
|---|---|---|
| Approval-Team Member Medical<br>Affairs | | 18 May 2016 11:33 CEST |
| Author-Trial Statistician | | 19 May 2016 20:43 CEST |
| Approval- Safety Evaluation<br>Therapeutic Area | | 20 May 2016 12:55 CEST |
| Approval-Medical | | 25 May 2016 10:22 CEST |
| Approval-Therapeutic Area | | 30 May 2016 11:53 CEST |

**Boehringer Ingelheim Document Number:** c09057375 **Technical Version Number:**1.0

#### (Continued) Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|----------------------|-----------|-------------|
|----------------------|-----------|-------------|